CLINICAL TRIAL: NCT00000611
Title: Women's Health Initiative (WHI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); National Cancer Institute (NCI) (NIH); National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 114
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2006-01

CONDITIONS: Bone Diseases; Breast Neoplasms; Cardiovascular Diseases; Colonic Neoplasms; Coronary Disease; Heart Diseases; Myocardial Ischemia; Osteoporosis; Postmenopause
MeSH Terms: conditions — Bone Diseases; Breast Neoplasms; Cardiovascular Diseases; Colonic Neoplasms; Coronary Disease; Heart Diseases; Myocardial Ischemia; Osteoporosis | interventions — Hormone Replacement Therapy; Estrogens; Progestins; Estrogen Replacement Therapy; Diet, Fat-Restricted; Calcium; Vitamin D; Dietary Supplements

INTERVENTIONS:
Drug: hormone replacement therapy
Drug: estrogens
Drug: progestins
Drug: estrogen replacement therapy
Behavioral: diet, fat-restricted
Drug: calcium
Drug: vitamin D
Behavioral: dietary supplements

SUMMARY:
To address cardiovascular disease, cancer, and osteoporosis, the most common causes of death, disability, and impaired quality of life in postmenopausal women. The three major components of the WHI are: a randomized controlled clinical trial of hormone replacement therapy (HRT), dietary modification (DM), and calcium/vitamin D supplementation (CaD); an observational study (OS); and a community prevention study (CPS). On October 1, 1997, administration of the WHI was transferred to the NHLBI where it is conducted as a consortium effort led by the NHLBI in cooperation with the National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS), the National Cancer Institute (NCI), and the National Institute on Aging (NIA).

DETAILED DESCRIPTION:
BACKGROUND:

Prior to 1991, little research had focused on health issues unique to, or more common for, women. This was especially the case for studies of chronic diseases and their prevention in mature women. These conditions (coronary heart disease, cancer, and osteoporosis) are the leading causes of impairment of quality of life, morbidity, and mortality in post-menopausal United States women. The WHI, mandated by Congress, was established in 1991 by the National Institutes of Health and located in the Office of the Director (OD). The Clinical Coordinating Center for the clinical trial/observational study was funded in September 1992 and the 16 Vanguard Clinical Centers were funded in March 1993. The initial protocol was developed jointly by the Clinical Coordinating Center and the Program Office and was reviewed and approved by the Investigators Committee on April 20, 1993. Additional clinical centers were funded in 1994.

On October 1, 1997, administration of the WHI was transferred to the NHLBI where it is conducted as a consortium effort led by the NHLBI in cooperation with the National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS), the National Cancer Institute (NCI), and the National Institute on Aging (NIA).

DESIGN NARRATIVE:

As has been described in the objective, the WHI has three major components: a randomized controlled clinical trial, an observational study, and a study of community approaches to developing healthful behaviors. Recruitment for the WHI began in September 1993 and ended in December 1998. Six clinical centers completed recruitment in January 1997. The remaining 34 centers completed recruitment in December 1998.

CLINICAL TRIAL COMPONENT

The clinical trial component consists of three subtrials: the hormone replacement trial, the dietary modification trial, and the calcium /vitamin D supplementation trial. Approximately 27,500 women aged 50 to 79 are participating in the HRT, which tests whether long-term HRT reduces coronary heart disease and fractures without increasing breast cancer risk. Women with a uterus were randomized to receive either estrogen plus progestin or a placebo. Progestin was added to protect women with a uterus from endometrial cancer. Women who have had a hysterectomy were randomized to receive either estrogen alone or a placebo. The estrogen plus progestin trial was stopped early on July 8, 2002 after an average follow-up of 5.2 years on the recommendation of the Data and Safety Monitoring Board. The estrogen alone study continued unchanged until March 2, 2004 when the NIH instructed participants to stop taking their study pills and to begin the follow-up phase of the study. . Participants in the estrogen alone study will be followed for eight to 12 years and have clinic visits every six months to assure safety and assess their health.

The dietary modification trial component studies the effect of a low-fat, high fruit, vegetable and grain diet on breast cancer, colorectal cancer and heart disease in 48,000 postmenopausal women. Participants are randomized to a comparison group which maintains usual dietary habits or to a dietary change group. Women in the dietary change group decrease their fat intake to 20 percent of total daily calories, increase fruit and vegetable consumption to five or more servings per day, and increase grains to six or more servings per day. Additionally, they monitor their food intake and attend nutrition group meetings to learn more about changing their diets in the first year. Thereafter they attend four meetings per year.

The calcium/vitamin D supplementation subtrial tests whether calcium and vitamin D supplements reduce the risk of hip and other fractures and colorectal cancer in postmenopausal women. Women in the hormone replacement therapy and the dietary modification trials are encouraged to join the calcium/vitamin D supplementation study. Approximately 45,000 postmenopausal women are randomized into one of two study groups. One group was randomly assigned to receive 1,000 mg of elemental calcium (as calcium carbonate) and 400 International Units of vitamin D₃daily. The second group received a matching placebo.

Women already taking calcium supplements can continue to take them. Participants will be followed for eight to 11 years and contacted by their clinical center every six months to assure their safety and assess their health.

Total number of trial participants in all three subtrials is 68,135.

OBSERVATIONAL STUDY

The several goals of the study include: to give reliable estimates of extent to which known risk factors predict heart disease, cancers, and fractures; to identify new risk factors for these and other diseases in women; to compare risk factors, presence of disease at the start of the study and new occurrences of disease during the WHI in all study components; and to create a future resource to identify biological indicators of disease, especially substances and factors found in blood. The study enrolled 93,726 postmenopausal women and will track them for an average of nine years. Participants fill out periodic health forms and visit the clinic three years after enrollment. They take no medication and do not change their health habits.

COMMUNITY PREVENTION STUDY

The community prevention study consists of 12 separate studies conducted at eight of the Centers for Disease Control and Prevention's (CDC) University-based Prevention Research Centers through a cooperative agreement between NIH and CDC. The 12 studies began in October 1995 and continue for an additional five years. The collaboration supports health promotion and disease prevention research and demonstration projects that are community-based and focus on healthy behaviors that prevent the major causes of death and disability and that promote health practices that lead to more effective public health interventions. Each project provides research dissemination and translation of findings into community interventions. Topics under study include: attitudes towards hysterectomy, oophorectomy, and surgical menopause among African Americans; reducing cardiovascular disease risk among Black women; environmental and policy interventions to increase physical activity among minority women ages 40 to 75; peer support intervention for cardiovascular disease risk among African American women, aged 40 and older; assessing the effectiveness of a brief medical-provider educational intervention for osteoporosis in minority women aged 40 and older; improving the delivery of diabetes care to women in minority groups; and assessment of moderate physical activity among women.

ELIGIBILITY:
Postmenopausal women ages 50 to 79.

Ages: 50 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Primary Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ross Prentice — Fred Hutchinson Cancer Center

REFERENCES:
- [Background] Rossouw JE, Hurd S. The Women's Health Initiative: recruitment complete--looking back and looking forward. J Womens Health. 1999 Jan-Feb;8(1):3-5. doi: 10.1089/jwh.1999.8.3. No abstract available. PMID 10094073
- [Background] Design of the Women's Health Initiative clinical trial and observational study. The Women's Health Initiative Study Group. Control Clin Trials. 1998 Feb;19(1):61-109. doi: 10.1016/s0197-2456(97)00078-0. PMID 9492970
- [Background] Patterson RE, Kristal AR, Tinker LF, Carter RA, Bolton MP, Agurs-Collins T. Measurement characteristics of the Women's Health Initiative food frequency questionnaire. Ann Epidemiol. 1999 Apr;9(3):178-87. doi: 10.1016/s1047-2797(98)00055-6. PMID 10192650
- [Background] McGowan JA, Pottern L. Commentary on the Women's Health Initiative. Maturitas. 2000 Feb 15;34(2):109-12. doi: 10.1016/s0378-5122(99)00109-7. PMID 10714904
- [Background] Wassertheil-Smoller S, Anderson G, Psaty BM, Black HR, Manson J, Wong N, Francis J, Grimm R, Kotchen T, Langer R, Lasser N. Hypertension and its treatment in postmenopausal women: baseline data from the Women's Health Initiative. Hypertension. 2000 Nov;36(5):780-9. doi: 10.1161/01.hyp.36.5.780. PMID 11082143
- [Background] Wilcox S, Shumaker SA, Bowen DJ, Naughton MJ, Rosal MC, Ludlam SE, Dugan E, Hunt JR, Stevens S. Promoting adherence and retention to clinical trials in special populations: a women's health initiative workshop. Control Clin Trials. 2001 Jun;22(3):279-89. doi: 10.1016/s0197-2456(00)00130-6. PMID 11384790
- [Background] Gottesman R. Medical care for minors without parental consent. Child Today. 1975 Mar-Apr;4(2):30-1. No abstract available. PMID 1116413
- [Background] Hsia J, Kemper E, Sofaer S, Bowen D, Kiefe CI, Zapka J, Mason E, Lillington L, Limacher M. Is insurance a more important determinant of healthcare access than perceived health? Evidence from the Women's Health Initiative. J Womens Health Gend Based Med. 2000 Oct;9(8):881-9. doi: 10.1089/152460900750020919. PMID 11074954
- [Background] Valanis BG, Bowen DJ, Bassford T, Whitlock E, Charney P, Carter RA. Sexual orientation and health: comparisons in the women's health initiative sample. Arch Fam Med. 2000 Sep-Oct;9(9):843-53. doi: 10.1001/archfami.9.9.843. PMID 11031391
- [Background] Hsia J, Kemper E, Kiefe C, Zapka J, Sofaer S, Pettinger M, Bowen D, Limacher M, Lillington L, Mason E. The importance of health insurance as a determinant of cancer screening: evidence from the Women's Health Initiative. Prev Med. 2000 Sep;31(3):261-70. doi: 10.1006/pmed.2000.0697. PMID 10964640
- [Background] Larkey LK, Staten LK, Ritenbaugh C, Hall RA, Buller DB, Bassford T, Altimari BR. Recruitment of Hispanic women to the Women's Health Initiative. the case of Embajadoras in Arizona. Control Clin Trials. 2002 Jun;23(3):289-98. doi: 10.1016/s0197-2456(02)00190-3. PMID 12057880
- [Background] Tinker LF, Perri MG, Patterson RE, Bowen DJ, McIntosh M, Parker LM, Sevick MA, Wodarski LA. The effects of physical and emotional status on adherence to a low-fat dietary pattern in the Women's Health Initiative. J Am Diet Assoc. 2002 Jun;102(6):789-800, 888. doi: 10.1016/s0002-8223(02)90178-1. PMID 12067044
- [Background] Hendrix SL, Clark A, Nygaard I, Aragaki A, Barnabei V, McTiernan A. Pelvic organ prolapse in the Women's Health Initiative: gravity and gravidity. Am J Obstet Gynecol. 2002 Jun;186(6):1160-6. doi: 10.1067/mob.2002.123819. PMID 12066091
- [Background] Rossouw JE, Anderson GL, Prentice RL, LaCroix AZ, Kooperberg C, Stefanick ML, Jackson RD, Beresford SA, Howard BV, Johnson KC, Kotchen JM, Ockene J; Writing Group for the Women's Health Initiative Investigators. Risks and benefits of estrogen plus progestin in healthy postmenopausal women: principal results From the Women's Health Initiative randomized controlled trial. JAMA. 2002 Jul 17;288(3):321-33. doi: 10.1001/jama.288.3.321. PMID 12117397
- [Background] Fletcher SW, Colditz GA. Failure of estrogen plus progestin therapy for prevention. JAMA. 2002 Jul 17;288(3):366-8. doi: 10.1001/jama.288.3.366. No abstract available. PMID 12117403
- [Background] Pradhan AD, Manson JE, Rossouw JE, Siscovick DS, Mouton CP, Rifai N, Wallace RB, Jackson RD, Pettinger MB, Ridker PM. Inflammatory biomarkers, hormone replacement therapy, and incident coronary heart disease: prospective analysis from the Women's Health Initiative observational study. JAMA. 2002 Aug 28;288(8):980-7. doi: 10.1001/jama.288.8.980. PMID 12190368
- [Background] Manson JE, Greenland P, LaCroix AZ, Stefanick ML, Mouton CP, Oberman A, Perri MG, Sheps DS, Pettinger MB, Siscovick DS. Walking compared with vigorous exercise for the prevention of cardiovascular events in women. N Engl J Med. 2002 Sep 5;347(10):716-25. doi: 10.1056/NEJMoa021067. PMID 12213942
- [Background] Shikany JM, Patterson RE, Agurs-Collins T, Anderson G. Antioxidant supplement use in Women's Health Initiative participants. Prev Med. 2003 Mar;36(3):379-87. doi: 10.1016/s0091-7435(02)00050-6. PMID 12634029
- [Background] Hays J, Ockene JK, Brunner RL, Kotchen JM, Manson JE, Patterson RE, Aragaki AK, Shumaker SA, Brzyski RG, LaCroix AZ, Granek IA, Valanis BG; Women's Health Initiative Investigators. Effects of estrogen plus progestin on health-related quality of life. N Engl J Med. 2003 May 8;348(19):1839-54. doi: 10.1056/NEJMoa030311. Epub 2003 Mar 17. PMID 12642637
- [Background] Rapp SR, Espeland MA, Shumaker SA, Henderson VW, Brunner RL, Manson JE, Gass ML, Stefanick ML, Lane DS, Hays J, Johnson KC, Coker LH, Dailey M, Bowen D; WHIMS Investigators. Effect of estrogen plus progestin on global cognitive function in postmenopausal women: the Women's Health Initiative Memory Study: a randomized controlled trial. JAMA. 2003 May 28;289(20):2663-72. doi: 10.1001/jama.289.20.2663. PMID 12771113
- [Background] Shumaker SA, Legault C, Rapp SR, Thal L, Wallace RB, Ockene JK, Hendrix SL, Jones BN 3rd, Assaf AR, Jackson RD, Kotchen JM, Wassertheil-Smoller S, Wactawski-Wende J; WHIMS Investigators. Estrogen plus progestin and the incidence of dementia and mild cognitive impairment in postmenopausal women: the Women's Health Initiative Memory Study: a randomized controlled trial. JAMA. 2003 May 28;289(20):2651-62. doi: 10.1001/jama.289.20.2651. PMID 12771112
- [Background] Wassertheil-Smoller S, Hendrix SL, Limacher M, Heiss G, Kooperberg C, Baird A, Kotchen T, Curb JD, Black H, Rossouw JE, Aragaki A, Safford M, Stein E, Laowattana S, Mysiw WJ; WHI Investigators. Effect of estrogen plus progestin on stroke in postmenopausal women: the Women's Health Initiative: a randomized trial. JAMA. 2003 May 28;289(20):2673-84. doi: 10.1001/jama.289.20.2673. PMID 12771114
- [Background] Chlebowski RT, Hendrix SL, Langer RD, Stefanick ML, Gass M, Lane D, Rodabough RJ, Gilligan MA, Cyr MG, Thomson CA, Khandekar J, Petrovitch H, McTiernan A; WHI Investigators. Influence of estrogen plus progestin on breast cancer and mammography in healthy postmenopausal women: the Women's Health Initiative Randomized Trial. JAMA. 2003 Jun 25;289(24):3243-53. doi: 10.1001/jama.289.24.3243. PMID 12824205
- [Background] Gann PH, Morrow M. Combined hormone therapy and breast cancer: a single-edged sword. JAMA. 2003 Jun 25;289(24):3304-6. doi: 10.1001/jama.289.24.3304. No abstract available. PMID 12824214
- [Background] Jackson M, Berman N, Huber M, Snetselaar L, Granek I, Boe K, Milas C, Spivak J, Chlebowski RT. Research staff turnover and participant adherence in the Women's Health Initiative. Control Clin Trials. 2003 Aug;24(4):422-35. doi: 10.1016/s0197-2456(03)00027-8. PMID 12865036
- [Background] Howard BV, Criqui MH, Curb JD, Rodabough R, Safford MM, Santoro N, Wilson AC, Wylie-Rosett J. Risk factor clustering in the insulin resistance syndrome and its relationship to cardiovascular disease in postmenopausal white, black, hispanic, and Asian/Pacific Islander women. Metabolism. 2003 Mar;52(3):362-71. doi: 10.1053/meta.2003.50057. PMID 12647277
- [Background] Hsia J, Barad D, Margolis K, Rodabough R, McGovern PG, Limacher MC, Oberman A, Smoller S; Women's Health Initiative Research Group. Usefulness of prior hysterectomy as an independent predictor of Framingham risk score (The Women's Health Initiative). Am J Cardiol. 2003 Aug 1;92(3):264-9. doi: 10.1016/s0002-9149(03)00621-0. PMID 12888128
- [Background] LaCroix AZ, Cauley JA, Pettinger M, Hsia J, Bauer DC, McGowan J, Chen Z, Lewis CE, McNeeley SG, Passaro MD, Jackson RD. Statin use, clinical fracture, and bone density in postmenopausal women: results from the Women's Health Initiative Observational Study. Ann Intern Med. 2003 Jul 15;139(2):97-104. doi: 10.7326/0003-4819-139-2-200307150-00009. PMID 12859159
- [Background] Cauley JA, Robbins J, Chen Z, Cummings SR, Jackson RD, LaCroix AZ, LeBoff M, Lewis CE, McGowan J, Neuner J, Pettinger M, Stefanick ML, Wactawski-Wende J, Watts NB; Women's Health Initiative Investigators. Effects of estrogen plus progestin on risk of fracture and bone mineral density: the Women's Health Initiative randomized trial. JAMA. 2003 Oct 1;290(13):1729-38. doi: 10.1001/jama.290.13.1729. PMID 14519707
- [Background] Anderson GL, Judd HL, Kaunitz AM, Barad DH, Beresford SA, Pettinger M, Liu J, McNeeley SG, Lopez AM; Women's Health Initiative Investigators. Effects of estrogen plus progestin on gynecologic cancers and associated diagnostic procedures: the Women's Health Initiative randomized trial. JAMA. 2003 Oct 1;290(13):1739-48. doi: 10.1001/jama.290.13.1739. PMID 14519708
- [Background] Chen Z, Pettinger MB, Ritenbaugh C, LaCroix AZ, Robbins J, Caan BJ, Barad DH, Hakim IA. Habitual tea consumption and risk of osteoporosis: a prospective study in the women's health initiative observational cohort. Am J Epidemiol. 2003 Oct 15;158(8):772-81. doi: 10.1093/aje/kwg214. PMID 14561667
- [Background] Hsia J, Criqui MH, Rodabough RJ, Langer RD, Resnick HE, Phillips LS, Allison M, Bonds DE, Masaki K, Caralis P, Kotchen JM; Women's Health Initiative Investigators. Estrogen plus progestin and the risk of peripheral arterial disease: the Women's Health Initiative. Circulation. 2004 Feb 10;109(5):620-6. doi: 10.1161/01.CIR.0000115309.63979.92. PMID 14769684
- [Background] Chlebowski RT, Wactawski-Wende J, Ritenbaugh C, Hubbell FA, Ascensao J, Rodabough RJ, Rosenberg CA, Taylor VM, Harris R, Chen C, Adams-Campbell LL, White E; Women's Health Initiative Investigators. Estrogen plus progestin and colorectal cancer in postmenopausal women. N Engl J Med. 2004 Mar 4;350(10):991-1004. doi: 10.1056/NEJMoa032071. PMID 14999111
- [Background] Hebert JR, Patterson RE, Gorfine M, Ebbeling CB, St Jeor ST, Chlebowski RT. Differences between estimated caloric requirements and self-reported caloric intake in the women's health initiative. Ann Epidemiol. 2003 Oct;13(9):629-37. doi: 10.1016/S1047-2797(03)00051-6. PMID 14732302
- [Background] Ritenbaugh C, Patterson RE, Chlebowski RT, Caan B, Fels-Tinker L, Howard B, Ockene J. The Women's Health Initiative Dietary Modification trial: overview and baseline characteristics of participants. Ann Epidemiol. 2003 Oct;13(9 Suppl):S87-97. doi: 10.1016/s1047-2797(03)00044-9. No abstract available. PMID 14575941
- [Background] Harris RE, Chlebowski RT, Jackson RD, Frid DJ, Ascenseo JL, Anderson G, Loar A, Rodabough RJ, White E, McTiernan A; Women's Health Initiative. Breast cancer and nonsteroidal anti-inflammatory drugs: prospective results from the Women's Health Initiative. Cancer Res. 2003 Sep 15;63(18):6096-101. PMID 14522941
- [Background] Morimoto LM, White E, Chen Z, Chlebowski RT, Hays J, Kuller L, Lopez AM, Manson J, Margolis KL, Muti PC, Stefanick ML, McTiernan A. Obesity, body size, and risk of postmenopausal breast cancer: the Women's Health Initiative (United States). Cancer Causes Control. 2002 Oct;13(8):741-51. doi: 10.1023/a:1020239211145. PMID 12420953
- [Background] Hsia J, Aragaki A, Bloch M, LaCroix AZ, Wallace R; WHI Investigators. Predictors of angina pectoris versus myocardial infarction from the Women's Health Initiative Observational Study. Am J Cardiol. 2004 Mar 15;93(6):673-8. doi: 10.1016/j.amjcard.2003.12.002. PMID 15019867
- [Background] Khurana C, Rosenbaum CG, Howard BV, Adams-Campbell LL, Detrano RC, Klouj A, Hsia J. Coronary artery calcification in black women and white women. Am Heart J. 2003 Apr;145(4):724-9. doi: 10.1067/mhj.2003.99. PMID 12679771
- [Background] Anderson GL, Limacher M, Assaf AR, Bassford T, Beresford SA, Black H, Bonds D, Brunner R, Brzyski R, Caan B, Chlebowski R, Curb D, Gass M, Hays J, Heiss G, Hendrix S, Howard BV, Hsia J, Hubbell A, Jackson R, Johnson KC, Judd H, Kotchen JM, Kuller L, LaCroix AZ, Lane D, Langer RD, Lasser N, Lewis CE, Manson J, Margolis K, Ockene J, O'Sullivan MJ, Phillips L, Prentice RL, Ritenbaugh C, Robbins J, Rossouw JE, Sarto G, Stefanick ML, Van Horn L, Wactawski-Wende J, Wallace R, Wassertheil-Smoller S; Women's Health Initiative Steering Committee. Effects of conjugated equine estrogen in postmenopausal women with hysterectomy: the Women's Health Initiative randomized controlled trial. JAMA. 2004 Apr 14;291(14):1701-12. doi: 10.1001/jama.291.14.1701. PMID 15082697
- [Background] Hulley SB, Grady D. The WHI estrogen-alone trial--do things look any better? JAMA. 2004 Apr 14;291(14):1769-71. doi: 10.1001/jama.291.14.1769. No abstract available. PMID 15082705
- [Background] Espeland MA, Rapp SR, Shumaker SA, Brunner R, Manson JE, Sherwin BB, Hsia J, Margolis KL, Hogan PE, Wallace R, Dailey M, Freeman R, Hays J; Women's Health Initiative Memory Study. Conjugated equine estrogens and global cognitive function in postmenopausal women: Women's Health Initiative Memory Study. JAMA. 2004 Jun 23;291(24):2959-68. doi: 10.1001/jama.291.24.2959. PMID 15213207
- [Background] Shumaker SA, Legault C, Kuller L, Rapp SR, Thal L, Lane DS, Fillit H, Stefanick ML, Hendrix SL, Lewis CE, Masaki K, Coker LH; Women's Health Initiative Memory Study. Conjugated equine estrogens and incidence of probable dementia and mild cognitive impairment in postmenopausal women: Women's Health Initiative Memory Study. JAMA. 2004 Jun 23;291(24):2947-58. doi: 10.1001/jama.291.24.2947. PMID 15213206
- [Background] Schneider LS. Estrogen and dementia: insights from the Women's Health Initiative Memory Study. JAMA. 2004 Jun 23;291(24):3005-7. doi: 10.1001/jama.291.24.3005. No abstract available. PMID 15213214
- [Background] Pradhan AD, LaCroix AZ, Langer RD, Trevisan M, Lewis CE, Hsia JA, Oberman A, Kotchen JM, Ridker PM. Tissue plasminogen activator antigen and D-dimer as markers for atherothrombotic risk among healthy postmenopausal women. Circulation. 2004 Jul 20;110(3):292-300. doi: 10.1161/01.CIR.0000134965.73212.A6. Epub 2004 Jul 6. PMID 15238458
- [Background] Fouad MN, Corbie-Smith G, Curb D, Howard BV, Mouton C, Simon M, Talavera G, Thompson J, Wang CY, White C, Young R. Special populations recruitment for the Women's Health Initiative: successes and limitations. Control Clin Trials. 2004 Aug;25(4):335-52. doi: 10.1016/j.cct.2004.03.005. PMID 15296809
- [Background] Margolis KL, Bonds DE, Rodabough RJ, Tinker L, Phillips LS, Allen C, Bassford T, Burke G, Torrens J, Howard BV; Women's Health Initiative Investigators. Effect of oestrogen plus progestin on the incidence of diabetes in postmenopausal women: results from the Women's Health Initiative Hormone Trial. Diabetologia. 2004 Jul;47(7):1175-1187. doi: 10.1007/s00125-004-1448-x. Epub 2004 Jul 14. PMID 15252707
- [Background] Naftolin F, Taylor HS, Karas R, Brinton E, Newman I, Clarkson TB, Mendelsohn M, Lobo RA, Judelson DR, Nachtigall LE, Heward CB, Hecht H, Jaff MR, Harman SM; Women's Health Initiative. The Women's Health Initiative could not have detected cardioprotective effects of starting hormone therapy during the menopausal transition. Fertil Steril. 2004 Jun;81(6):1498-501. doi: 10.1016/j.fertnstert.2004.02.095. PMID 15193467
- [Background] Chen Z, Kooperberg C, Pettinger MB, Bassford T, Cauley JA, LaCroix AZ, Lewis CE, Kipersztok S, Borne C, Jackson RD. Validity of self-report for fractures among a multiethnic cohort of postmenopausal women: results from the Women's Health Initiative observational study and clinical trials. Menopause. 2004 May-Jun;11(3):264-74. doi: 10.1097/01.gme.0000094210.15096.fd. PMID 15167305
- [Background] Women's Health Initiative Study Group. Dietary adherence in the Women's Health Initiative Dietary Modification Trial. J Am Diet Assoc. 2004 Apr;104(4):654-8. doi: 10.1016/j.jada.2004.01.014. PMID 15054353
- [Background] Cushman M, Kuller LH, Prentice R, Rodabough RJ, Psaty BM, Stafford RS, Sidney S, Rosendaal FR; Women's Health Initiative Investigators. Estrogen plus progestin and risk of venous thrombosis. JAMA. 2004 Oct 6;292(13):1573-80. doi: 10.1001/jama.292.13.1573. PMID 15467059
- [Background] Heckbert SR, Kooperberg C, Safford MM, Psaty BM, Hsia J, McTiernan A, Gaziano JM, Frishman WH, Curb JD. Comparison of self-report, hospital discharge codes, and adjudication of cardiovascular events in the Women's Health Initiative. Am J Epidemiol. 2004 Dec 15;160(12):1152-8. doi: 10.1093/aje/kwh314. PMID 15583367
- [Background] Wassertheil-Smoller S, Psaty B, Greenland P, Oberman A, Kotchen T, Mouton C, Black H, Aragaki A, Trevisan M. Association between cardiovascular outcomes and antihypertensive drug treatment in older women. JAMA. 2004 Dec 15;292(23):2849-59. doi: 10.1001/jama.292.23.2849. PMID 15598916
- [Background] Espeland MA, Gu L, Masaki KH, Langer RD, Coker LH, Stefanick ML, Ockene J, Rapp SR. Association between reported alcohol intake and cognition: results from the Women's Health Initiative Memory Study. Am J Epidemiol. 2005 Feb 1;161(3):228-38. doi: 10.1093/aje/kwi043. PMID 15671255
- [Background] Howard BV, Adams-Campbell L, Allen C, Black H, Passaro M, Rodabough RJ, Rodriguez BL, Safford M, Stevens VJ, Wagenknecht LE. Insulin resistance and weight gain in postmenopausal women of diverse ethnic groups. Int J Obes Relat Metab Disord. 2004 Aug;28(8):1039-47. doi: 10.1038/sj.ijo.0802645. PMID 15254486
- [Background] Hendrix SL, Cochrane BB, Nygaard IE, Handa VL, Barnabei VM, Iglesia C, Aragaki A, Naughton MJ, Wallace RB, McNeeley SG. Effects of estrogen with and without progestin on urinary incontinence. JAMA. 2005 Feb 23;293(8):935-48. doi: 10.1001/jama.293.8.935. PMID 15728164
- [Background] Curb JD, McTiernan A, Heckbert SR, Kooperberg C, Stanford J, Nevitt M, Johnson KC, Proulx-Burns L, Pastore L, Criqui M, Daugherty S; WHI Morbidity and Mortality Committee. Outcomes ascertainment and adjudication methods in the Women's Health Initiative. Ann Epidemiol. 2003 Oct;13(9 Suppl):S122-8. doi: 10.1016/s1047-2797(03)00048-6. No abstract available. PMID 14575944
- [Background] Hsia J, Wu L, Allen C, Oberman A, Lawson WE, Torrens J, Safford M, Limacher MC, Howard BV; Women's Health Initiative Research Group. Physical activity and diabetes risk in postmenopausal women. Am J Prev Med. 2005 Jan;28(1):19-25. doi: 10.1016/j.amepre.2004.09.012. PMID 15626551
- [Background] Cirillo DJ, Wallace RB, Rodabough RJ, Greenland P, LaCroix AZ, Limacher MC, Larson JC. Effect of estrogen therapy on gallbladder disease. JAMA. 2005 Jan 19;293(3):330-9. doi: 10.1001/jama.293.3.330. PMID 15657326
- [Background] Margolis KL, Manson JE, Greenland P, Rodabough RJ, Bray PF, Safford M, Grimm RH Jr, Howard BV, Assaf AR, Prentice R; Women's Health Initiative Research Group. Leukocyte count as a predictor of cardiovascular events and mortality in postmenopausal women: the Women's Health Initiative Observational Study. Arch Intern Med. 2005 Mar 14;165(5):500-8. doi: 10.1001/archinte.165.5.500. PMID 15767524
- [Background] Howard BV, Kuller L, Langer R, Manson JE, Allen C, Assaf A, Cochrane BB, Larson JC, Lasser N, Rainford M, Van Horn L, Stefanick ML, Trevisan M; Women's Health Initiative. Risk of cardiovascular disease by hysterectomy status, with and without oophorectomy: the Women's Health Initiative Observational Study. Circulation. 2005 Mar 29;111(12):1462-70. doi: 10.1161/01.CIR.0000159344.21672.FD. Epub 2005 Mar 21. PMID 15781742
- [Background] Langer RD, Pradhan AD, Lewis CE, Manson JE, Rossouw JE, Hendrix SL, LaCroix AZ, Ridker PM. Baseline associations between postmenopausal hormone therapy and inflammatory, haemostatic, and lipid biomarkers of coronary heart disease. The Women's Health Initiative Observational Study. Thromb Haemost. 2005 Jun;93(6):1108-16. doi: 10.1160/TH04-09-0608. PMID 15968396
- [Background] Ockene JK, Barad DH, Cochrane BB, Larson JC, Gass M, Wassertheil-Smoller S, Manson JE, Barnabei VM, Lane DS, Brzyski RG, Rosal MC, Wylie-Rosett J, Hays J. Symptom experience after discontinuing use of estrogen plus progestin. JAMA. 2005 Jul 13;294(2):183-93. doi: 10.1001/jama.294.2.183. PMID 16014592
- [Background] Chen Z, Maricic M, Bassford TL, Pettinger M, Ritenbaugh C, Lopez AM, Barad DH, Gass M, Leboff MS. Fracture risk among breast cancer survivors: results from the Women's Health Initiative Observational Study. Arch Intern Med. 2005 Mar 14;165(5):552-8. doi: 10.1001/archinte.165.5.552. PMID 15767532
- [Background] Woods NF, LaCroix AZ, Gray SL, Aragaki A, Cochrane BB, Brunner RL, Masaki K, Murray A, Newman AB; Women's Health Initiative. Frailty: emergence and consequences in women aged 65 and older in the Women's Health Initiative Observational Study. J Am Geriatr Soc. 2005 Aug;53(8):1321-30. doi: 10.1111/j.1532-5415.2005.53405.x. PMID 16078957
- [Background] Michael YL, Perrin N, Bowen D, Cochrane BB, Wisdom JP, Brzyski R, Ritenbaugh C. Expression and ambivalence over expression of negative emotion:psychometric analysis in the Women's Health Initiative. J Women Aging. 2005;17(1-2):5-18. doi: 10.1300/J074v17n01_02. PMID 15914416
- [Background] Barnabei VM, Cochrane BB, Aragaki AK, Nygaard I, Williams RS, McGovern PG, Young RL, Wells EC, O'Sullivan MJ, Chen B, Schenken R, Johnson SR; Women's Health Initiative Investigators. Menopausal symptoms and treatment-related effects of estrogen and progestin in the Women's Health Initiative. Obstet Gynecol. 2005 May;105(5 Pt 1):1063-73. doi: 10.1097/01.AOG.0000158120.47542.18. PMID 15863546
- [Background] Stefanick ML, Prentice RL, Anderson G, Gass M, Manson JE, Hendrix SL, Vista-Deck D, McNeeley G; Women's Health Initiative Steering Committee. Reanalysis of the Women's Health Initiative oral contraceptive data reveals no evidence of delayed cardiovascular benefit. Fertil Steril. 2005 Apr;83(4):853-4. doi: 10.1016/j.fertnstert.2005.01.084. PMID 15820789
- [Background] Brunner RL, Gass M, Aragaki A, Hays J, Granek I, Woods N, Mason E, Brzyski R, Ockene J, Assaf A, LaCroix A, Matthews K, Wallace R; Women's Health Initiative Investigators. Effects of conjugated equine estrogen on health-related quality of life in postmenopausal women with hysterectomy: results from the Women's Health Initiative Randomized Clinical Trial. Arch Intern Med. 2005 Sep 26;165(17):1976-86. doi: 10.1001/archinte.165.17.1976. PMID 16186467
- [Background] Wampler NS, Chen Z, Jacobsen C, Henderson JA, Howard BV, Rossouw JE. Bone mineral density of American Indian and Alaska Native women compared with non-Hispanic white women: results from the Women's Health Initiative Study. Menopause. 2005 Sep-Oct;12(5):536-44. doi: 10.1097/01.gme.0000182161.88939.f0. Epub 2005 Sep 1. PMID 16145307
- [Background] Prentice RL, Langer R, Stefanick ML, Howard BV, Pettinger M, Anderson G, Barad D, Curb JD, Kotchen J, Kuller L, Limacher M, Wactawski-Wende J; Women's Health Initiative Investigators. Combined postmenopausal hormone therapy and cardiovascular disease: toward resolving the discrepancy between observational studies and the Women's Health Initiative clinical trial. Am J Epidemiol. 2005 Sep 1;162(5):404-14. doi: 10.1093/aje/kwi223. Epub 2005 Jul 20. PMID 16033876
- [Background] Chen Z, Bassford T, Green SB, Cauley JA, Jackson RD, LaCroix AZ, Leboff M, Stefanick ML, Margolis KL. Postmenopausal hormone therapy and body composition--a substudy of the estrogen plus progestin trial of the Women's Health Initiative. Am J Clin Nutr. 2005 Sep;82(3):651-6. doi: 10.1093/ajcn.82.3.651. PMID 16155280
- [Background] Wolf RL, Cauley JA, Pettinger M, Jackson R, Lacroix A, Leboff MS, Lewis CE, Nevitt MC, Simon JA, Stone KL, Wactawski-Wende J. Lack of a relation between vitamin and mineral antioxidants and bone mineral density: results from the Women's Health Initiative. Am J Clin Nutr. 2005 Sep;82(3):581-8. doi: 10.1093/ajcn.82.3.581. PMID 16155271
- [Background] Barad D, Kooperberg C, Wactawski-Wende J, Liu J, Hendrix SL, Watts NB. Prior oral contraception and postmenopausal fracture: a Women's Health Initiative observational cohort study. Fertil Steril. 2005 Aug;84(2):374-83. doi: 10.1016/j.fertnstert.2005.01.132. PMID 16084878
- [Background] Howard BV, Manson JE, Stefanick ML, Beresford SA, Frank G, Jones B, Rodabough RJ, Snetselaar L, Thomson C, Tinker L, Vitolins M, Prentice R. Low-fat dietary pattern and weight change over 7 years: the Women's Health Initiative Dietary Modification Trial. JAMA. 2006 Jan 4;295(1):39-49. doi: 10.1001/jama.295.1.39. PMID 16391215
- [Background] Women's Health Initiative Steering Committee: Effects of Conjugated Equine Estrogen in Postmenopausal Women Having Undergone Hysterectomy: The Women's Health Initiative Randomized, Controlled Trials. Obstet Gynecol Surv, 59(8):599-600, 2004.
- [Result] Stefanick ML, Anderson GL, Margolis KL, Hendrix SL, Rodabough RJ, Paskett ED, Lane DS, Hubbell FA, Assaf AR, Sarto GE, Schenken RS, Yasmeen S, Lessin L, Chlebowski RT; WHI Investigators. Effects of conjugated equine estrogens on breast cancer and mammography screening in postmenopausal women with hysterectomy. JAMA. 2006 Apr 12;295(14):1647-57. doi: 10.1001/jama.295.14.1647. PMID 16609086
- [Result] Jackson RD, LaCroix AZ, Gass M, Wallace RB, Robbins J, Lewis CE, Bassford T, Beresford SA, Black HR, Blanchette P, Bonds DE, Brunner RL, Brzyski RG, Caan B, Cauley JA, Chlebowski RT, Cummings SR, Granek I, Hays J, Heiss G, Hendrix SL, Howard BV, Hsia J, Hubbell FA, Johnson KC, Judd H, Kotchen JM, Kuller LH, Langer RD, Lasser NL, Limacher MC, Ludlam S, Manson JE, Margolis KL, McGowan J, Ockene JK, O'Sullivan MJ, Phillips L, Prentice RL, Sarto GE, Stefanick ML, Van Horn L, Wactawski-Wende J, Whitlock E, Anderson GL, Assaf AR, Barad D; Women's Health Initiative Investigators. Calcium plus vitamin D supplementation and the risk of fractures. N Engl J Med. 2006 Feb 16;354(7):669-83. doi: 10.1056/NEJMoa055218. PMID 16481635
- [Result] Howard BV, Van Horn L, Hsia J, Manson JE, Stefanick ML, Wassertheil-Smoller S, Kuller LH, LaCroix AZ, Langer RD, Lasser NL, Lewis CE, Limacher MC, Margolis KL, Mysiw WJ, Ockene JK, Parker LM, Perri MG, Phillips L, Prentice RL, Robbins J, Rossouw JE, Sarto GE, Schatz IJ, Snetselaar LG, Stevens VJ, Tinker LF, Trevisan M, Vitolins MZ, Anderson GL, Assaf AR, Bassford T, Beresford SA, Black HR, Brunner RL, Brzyski RG, Caan B, Chlebowski RT, Gass M, Granek I, Greenland P, Hays J, Heber D, Heiss G, Hendrix SL, Hubbell FA, Johnson KC, Kotchen JM. Low-fat dietary pattern and risk of cardiovascular disease: the Women's Health Initiative Randomized Controlled Dietary Modification Trial. JAMA. 2006 Feb 8;295(6):655-66. doi: 10.1001/jama.295.6.655. PMID 16467234
- [Result] Beresford SA, Johnson KC, Ritenbaugh C, Lasser NL, Snetselaar LG, Black HR, Anderson GL, Assaf AR, Bassford T, Bowen D, Brunner RL, Brzyski RG, Caan B, Chlebowski RT, Gass M, Harrigan RC, Hays J, Heber D, Heiss G, Hendrix SL, Howard BV, Hsia J, Hubbell FA, Jackson RD, Kotchen JM, Kuller LH, LaCroix AZ, Lane DS, Langer RD, Lewis CE, Manson JE, Margolis KL, Mossavar-Rahmani Y, Ockene JK, Parker LM, Perri MG, Phillips L, Prentice RL, Robbins J, Rossouw JE, Sarto GE, Stefanick ML, Van Horn L, Vitolins MZ, Wactawski-Wende J, Wallace RB, Whitlock E. Low-fat dietary pattern and risk of colorectal cancer: the Women's Health Initiative Randomized Controlled Dietary Modification Trial. JAMA. 2006 Feb 8;295(6):643-54. doi: 10.1001/jama.295.6.643. PMID 16467233
- [Result] Prentice RL, Caan B, Chlebowski RT, Patterson R, Kuller LH, Ockene JK, Margolis KL, Limacher MC, Manson JE, Parker LM, Paskett E, Phillips L, Robbins J, Rossouw JE, Sarto GE, Shikany JM, Stefanick ML, Thomson CA, Van Horn L, Vitolins MZ, Wactawski-Wende J, Wallace RB, Wassertheil-Smoller S, Whitlock E, Yano K, Adams-Campbell L, Anderson GL, Assaf AR, Beresford SA, Black HR, Brunner RL, Brzyski RG, Ford L, Gass M, Hays J, Heber D, Heiss G, Hendrix SL, Hsia J, Hubbell FA, Jackson RD, Johnson KC, Kotchen JM, LaCroix AZ, Lane DS, Langer RD, Lasser NL, Henderson MM. Low-fat dietary pattern and risk of invasive breast cancer: the Women's Health Initiative Randomized Controlled Dietary Modification Trial. JAMA. 2006 Feb 8;295(6):629-42. doi: 10.1001/jama.295.6.629. PMID 16467232
- [Result] Yasmeen S, Romano PS, Pettinger M, Johnson SR, Hubbell FA, Lane DS, Hendrix SL. Incidence of cervical cytological abnormalities with aging in the women's health initiative: a randomized controlled trial. Obstet Gynecol. 2006 Aug;108(2):410-9. doi: 10.1097/01.AOG.0000225976.69396.fb. PMID 16880313
- [Derived] Prentice RL, Tinker LF, Neuhouser ML, Lampe JW, Raftery D, Gowda GN, Song X, Navarro SL, Huang Y, Vasan S, Orchard TS, Brasky TM, Manson JE, Zheng C. Biomarkers for dietary fatty acid densities among postmenopausal United States females derived using a habitual-diet human feeding study. Am J Clin Nutr. 2026 Jan 14:101197. doi: 10.1016/j.ajcnut.2026.101197. Online ahead of print. PMID 41544713
- [Derived] Zuraikat FM, Cheng B, Jelic S, Tasali E, Cespedes Feliciano EM, Saquib N, Shadyab AH, Titcomb TJ, Snetselaar LG, Hayden KM, Sanderlin AH, Molina-Henry DP, LeBlanc ES, St-Onge MP. Greater adherence to healthful dietary patterns is associated with lower insomnia risk in the Women's Health Initiative Observational Study. Sleep. 2026 Jan 13;49(1):zsaf316. doi: 10.1093/sleep/zsaf316. PMID 41065709
- [Derived] Johnson JJ, Ghosh S, Shaw PA, Neuhouser ML, Lampe JW, Tinker LF, Prentice RL, Tasevska N, Freedman LS, Boyer BB, Hopkins SE, Nash SH, Votruba SB, Krakoff J, O'Brien DM. The carbon isotope ratio of alanine is a biomarker of added sugar and sugar-sweetened beverage intakes: a pooled analysis of 4 studies. Am J Clin Nutr. 2025 Dec;122(6):1769-1777. doi: 10.1016/j.ajcnut.2025.09.049. Epub 2025 Oct 3. PMID 41047130
- [Derived] Rossouw JE, Aragaki AK, Manson JE, Szmuilowicz ED, Harrington LB, Johnson KC, Allison M, Haring B, Saquib N, Shadyab AH, Rexrode KM, Liu L, Mouton CP, LaCroix AZ. Menopausal Hormone Therapy and Cardiovascular Diseases in Women With Vasomotor Symptoms: A Secondary Analysis of the Women's Health Initiative Randomized Clinical Trials. JAMA Intern Med. 2025 Nov 1;185(11):1330-1339. doi: 10.1001/jamainternmed.2025.4510. PMID 40952729
- [Derived] Ezzat D, Uddin MM, Xue L, Pershad Y, Zhang S, Collins JM, Kitzman JO, Jaiswal S, Desai P, Kooperberg C, Bick AG, Natarajan P, Manson JE, Whitsel EA, Reiner AP, Honigberg MC. Clonal Hematopoiesis and Cardiovascular Outcomes in Older Women. J Am Coll Cardiol. 2025 Oct 14;86(15):1093-1106. doi: 10.1016/j.jacc.2025.07.058. Epub 2025 Aug 27. PMID 40864016
- [Derived] Baillie HT, Tinker LF, An P, Brasky TM, Liu S, Manson JE, Snetselaar L, Tabung FK, Lampe JW, Neuhouser ML. Dietary Supplement Use Is Associated with Select Serum Nutrient Biomarkers among Postmenopausal Women: Results from a Controlled Feeding Study. J Nutr. 2025 Aug;155(8):2745-2754. doi: 10.1016/j.tjnut.2025.06.003. Epub 2025 Jun 9. PMID 40499654
- [Derived] Thomson CA, Basen-Engquist K, Robles-Morales R, Roe DJ, Erdrich J, Trabert B, Saquib N, Cote ML, Qi L, Lane DS, Crane TE. Epidemiological Analysis of Obesity-related co-morbidities and mortality among post- menopausal women diagnosed with endometrial cancer: A Randomized Controlled Trial. Res Sq [Preprint]. 2025 Apr 8:rs.3.rs-6214415. doi: 10.21203/rs.3.rs-6214415/v1. PMID 40297687
- [Derived] Prentice RL, Aragaki AK, Zheng C, Manson JE, Tinker LF, Schoeller DA, Ravelli MN, Raftery D, Gowda GN, Navarro SL, Huang Y, Mossavar-Rahmani Y, Wallace RB, Johnson KC, Lampe JW, Neuhouser ML. Energy intake is associated with dietary macronutrient densities: inversely with protein and monounsaturated fat and positively with polyunsaturated fat and carbohydrate among postmenopausal females. Am J Clin Nutr. 2025 May;121(5):1165-1175. doi: 10.1016/j.ajcnut.2025.03.011. Epub 2025 Mar 13. PMID 40088973
- [Derived] Nudy M, Aragaki AK, Jiang X, Manson JE, Shadyab AH, Jung SY, Martin LW, Wild RA, Womack C, Mouton CP, Rossouw JE, Schnatz PF. Long-Term Changes to Cardiovascular Biomarkers After Hormone Therapy in the Women's Health Initiative Hormone Therapy Clinical Trials. Obstet Gynecol. 2025 Apr 1;145(4):357-367. doi: 10.1097/AOG.0000000000005862. Epub 2025 Feb 27. PMID 40014858
- [Derived] Cheng RK, Roberts MB, Bansal N, Reding K, Salahuddin T, Mamas M, LaMonte M, Shadyab AH, Franceschini N, Klein L, Manson JE, Eaton CB. Association of Kidney Function With Incident Heart Failure: An Analysis of the Women's Health Initiative. J Am Heart Assoc. 2025 Mar 4;14(5):e037051. doi: 10.1161/JAHA.124.037051. Epub 2025 Feb 25. PMID 39996449
- [Derived] Bea JW, Ochs-Balcom HM, Valencia CI, Chen Z, Blew RM, Lind KE, Caan BJ, Roe DJ, Rohan TE, Reeves KW, Manson JE, Ballinger T, Reding KW, Follis S, Ziller SG, Odegaard AO. Abdominal visceral and subcutaneous adipose tissue associations with postmenopausal breast cancer incidence. JNCI Cancer Spectr. 2025 Jan 3;9(1):pkaf007. doi: 10.1093/jncics/pkaf007. PMID 39847539
- [Derived] Chlebowski RT, Aragaki AK, Pan K, Haque R, Rohan TE, Song M, Wactawski-Wende J, Lane DS, Harris HR, Strickler H, Kauntiz AM, Runowicz CD. Menopausal Hormone Therapy and Ovarian and Endometrial Cancers: Long-Term Follow-Up of the Women's Health Initiative Randomized Trials. J Clin Oncol. 2024 Oct 20;42(30):3537-3549. doi: 10.1200/JCO.23.01918. Epub 2024 Aug 22. PMID 39173088
- [Derived] Dilek S, Figen Y, Merve G, Hatice EO, Seyma KT. Technology versus nostalgia; A randomized controlled trial of the effect of virtual reality and kaleidescop on pediatric pain, fear and anxiety management during immunization. J Pediatr Nurs. 2024 Sep-Oct;78:e383-e388. doi: 10.1016/j.pedn.2024.07.029. Epub 2024 Aug 1. PMID 39089900
- [Derived] Chlebowski RT, Aragaki AK, Pan K, Luo J, Rohan TE, Johnson KC, Wactawski-Wende J, Jung SY, Xiao Q, Lavasani S, Manson JE, Simon MS. Estrogen Plus Progestin and Colorectal Cancer: Long-Term Findings From the Women's Health Initiative Randomized Clinical Trial. J Clin Oncol. 2024 Oct 20;42(30):3530-3536. doi: 10.1200/JCO.23.02092. Epub 2024 Jul 19. PMID 39028918
- [Derived] Thomson CA, Aragaki AK, Prentice RL, Stefanick ML, Manson JE, Wactawski-Wende J, Watts NB, Van Horn L, Shikany JM, Rohan TE, Lane DS, Wild RA, Robles-Morales R, Shadyab AH, Saquib N, Cauley J. Long-Term Effect of Randomization to Calcium and Vitamin D Supplementation on Health in Older Women : Postintervention Follow-up of a Randomized Clinical Trial. Ann Intern Med. 2024 Apr;177(4):428-438. doi: 10.7326/M23-2598. Epub 2024 Mar 12. PMID 38467003
- [Derived] Prentice RL, Aragaki AK, Zheng C, Manson JE, Tinker LF, Ravelli MN, Mossavar-Rahmani Y, Wallace RB, Tooze JA, Johnson KC, Lampe JW, Neuhouser ML, Schoeller DA. Biomarker-assessed total energy intake and its cohort study association with all-cause mortality in postmenopausal females. Am J Clin Nutr. 2024 May;119(5):1329-1337. doi: 10.1016/j.ajcnut.2024.02.020. Epub 2024 Feb 29. PMID 38428741
- [Derived] Playdon MC, Tinker LF, Prentice RL, Loftfield E, Hayden KM, Van Horn L, Sampson JN, Stolzenberg-Solomon R, Lampe JW, Neuhouser ML, Moore SC. Measuring diet by metabolomics: a 14-d controlled feeding study of weighed food intake. Am J Clin Nutr. 2024 Feb;119(2):511-526. doi: 10.1016/j.ajcnut.2023.10.016. Epub 2023 Dec 29. PMID 38212160
- [Derived] Lara LA, Cartagena-Ramos D, Figueiredo JB, Rosa-E-Silva ACJ, Ferriani RA, Martins WP, Fuentealba-Torres M. Hormone therapy for sexual function in perimenopausal and postmenopausal women. Cochrane Database Syst Rev. 2023 Aug 24;8(8):CD009672. doi: 10.1002/14651858.CD009672.pub3. PMID 37619252
- [Derived] Prentice RL, Vasan S, Tinker LF, Neuhouser ML, Navarro SL, Raftery D, Gowda GN, Pettinger M, Aragaki AK, Lampe JW, Huang Y, Van Horn L, Manson JE, Wallace R, Mossavar-Rahmani Y, Wactawski-Wende J, Liu S, Snetselaar L, Howard BV, Chlebowski RT, Zheng C. Metabolomics-Based Biomarker for Dietary Fat and Associations with Chronic Disease Risk in Postmenopausal Women. J Nutr. 2023 Sep;153(9):2651-2662. doi: 10.1016/j.tjnut.2023.05.021. Epub 2023 May 26. PMID 37245660
- [Derived] Prentice RL, Vasan S, Tinker LF, Neuhouser ML, Navarro SL, Raftery D, Gowda GN, Pettinger M, Aragaki AK, Lampe JW, Huang Y, Van Horn L, Manson JE, Wallace RB, Mossavar-Rahmani Y, Wactawski-Wende J, Liu S, Snetselaar L, Howard BV, Chlebowski RT, Zheng C. Metabolomics Biomarkers for Fatty Acid Intake and Biomarker-Calibrated Fatty Acid Associations with Chronic Disease Risk in Postmenopausal Women. J Nutr. 2023 Sep;153(9):2663-2677. doi: 10.1016/j.tjnut.2023.05.003. Epub 2023 May 12. PMID 37178978
- [Derived] Prentice RL, Aragaki AK, Manson JE, Schoeller DA, Tinker LF, Mossavar-Rahmani Y, Wallace RB, LaMonte MJ, Tooze JA, Johnson KC, Lampe JW, Neuhouser ML. Total energy expenditure as assessed by doubly labeled water and all-cause mortality in a cohort of postmenopausal women. Am J Clin Nutr. 2023 May;117(5):955-963. doi: 10.1016/j.ajcnut.2023.02.023. Epub 2023 Mar 6. PMID 36889672
- [Derived] Neuhouser ML, Pettinger M, Tinker LF, Thomson C, Van Horn L, Haring B, Shikany JM, Stefanick ML, Prentice RL, Manson JE, Mossavar-Rahmani Y, Lampe JW. Associations of Biomarker-Calibrated Healthy Eating Index-2010 Scores with Chronic Disease Risk and Their Dependency on Energy Intake and Body Mass Index in Postmenopausal Women. J Nutr. 2023 Jan 14;152(12):2808-2817. doi: 10.1093/jn/nxac199. PMID 36040344
- [Derived] Pan K, Aragaki AK, Michael Y, Thomson CA, Snetselaar LG, Wactawski-Wende J, Garcia DO, Dieli-Conwright CM, Shadyab AH, Saquib N, Chlebowski RT. Long-term dietary intervention influence on physical activity in the Women's Health Initiative Dietary Modification randomized trial. Breast Cancer Res Treat. 2022 Aug;195(1):43-54. doi: 10.1007/s10549-022-06655-8. Epub 2022 Jul 12. PMID 35821536
- [Derived] Larson SR, Vasbinder AL, Reding KW, Leary PJ, Branch KR, Shadyab AH, Johnson KC, Haring B, Wallace R, Manson JE, Anderson G, Cheng RK. Histamine H2 Receptor Antagonists and Heart Failure Risk in Postmenopausal Women: The Women's Health Initiative. J Am Heart Assoc. 2022 Mar;11(5):e024270. doi: 10.1161/JAHA.121.024270. Epub 2022 Feb 22. PMID 35191329
- [Derived] Cene CW, Leng XI, Faraz K, Allison M, Breathett K, Bird C, Coday M, Corbie-Smith G, Foraker R, Ijioma NN, Rosal MC, Sealy-Jefferson S, Shippee TP, Kroenke CH. Social Isolation and Incident Heart Failure Hospitalization in Older Women: Women's Health Initiative Study Findings. J Am Heart Assoc. 2022 Mar;11(5):e022907. doi: 10.1161/JAHA.120.022907. Epub 2022 Feb 22. PMID 35189692
- [Derived] Tinker LF, Huang Y, Johnson KC, Carbone LD, Snetselaar L, Van Horn L, Manson JE, Liu S, Mossavar-Rahmani Y, Prentice RL, Lampe JW, Neuhouser ML. Estimating 24-Hour Urinary Excretion of Sodium and Potassium Is More Reliable from 24-Hour Urine Than Spot Urine Sample in a Feeding Study of US Older Postmenopausal Women. Curr Dev Nutr. 2021 Oct 12;5(11):nzab125. doi: 10.1093/cdn/nzab125. eCollection 2021 Nov. PMID 34761160
- [Derived] Pan K, Aragaki AK, Neuhouser ML, Simon MS, Luo J, Caan B, Snetselaar L, Mortimer JE, Manson JE, Kroenke C, Lane D, Reding K, Rohan TE, Chlebowski RT. Low-fat dietary pattern and breast cancer mortality by metabolic syndrome components: a secondary analysis of the Women's Health Initiative (WHI) randomised trial. Br J Cancer. 2021 Aug;125(3):372-379. doi: 10.1038/s41416-021-01379-w. Epub 2021 May 18. PMID 34006923
- [Derived] Prentice RL, Pettinger M, Neuhouser ML, Raftery D, Zheng C, Gowda GAN, Huang Y, Tinker LF, Howard BV, Manson JE, Wallace R, Mossavar-Rahmani Y, Johnson KC, Lampe JW. Biomarker-Calibrated Macronutrient Intake and Chronic Disease Risk among Postmenopausal Women. J Nutr. 2021 Aug 7;151(8):2330-2341. doi: 10.1093/jn/nxab091. PMID 33880504
- [Derived] Prentice RL, Howard BV, Van Horn L, Neuhouser ML, Anderson GL, Tinker LF, Lampe JW, Raftery D, Pettinger M, Aragaki AK, Thomson CA, Mossavar-Rahmani Y, Stefanick ML, Cauley JA, Rossouw JE, Manson JE, Chlebowski RT. Nutritional epidemiology and the Women's Health Initiative: a review. Am J Clin Nutr. 2021 May 8;113(5):1083-1092. doi: 10.1093/ajcn/nqab091. PMID 33876183
- [Derived] Flores M, Ruiz JM, Butler EA, Sbarra DA, Garcia DO, Kohler L, Crane TE, Corbie-Smith G, Benavente V, Kroenke CH, Saquib N, Thomson CA. Does the Hispanic Mortality Advantage Vary by Marital Status Among Postmenopausal Women in the Women's Health Initiative? Ann Behav Med. 2021 Jun 28;55(7):612-620. doi: 10.1093/abm/kaaa113. PMID 33449073
- [Derived] Hooper L, Martin N, Jimoh OF, Kirk C, Foster E, Abdelhamid AS. Reduction in saturated fat intake for cardiovascular disease. Cochrane Database Syst Rev. 2020 Aug 21;8(8):CD011737. doi: 10.1002/14651858.CD011737.pub3. PMID 32827219
- [Derived] Wang A, Zawadzki N, Hedlin H, LeBlanc E, Budrys N, Van Horn L, Gass M, Westphal L, Stefanick ML. Reproductive history and osteoarthritis in the Women's Health Initiative. Scand J Rheumatol. 2021 Jan;50(1):58-67. doi: 10.1080/03009742.2020.1751271. Epub 2020 Aug 6. PMID 32757806
- [Derived] Yun HY, Tinker LF, Neuhouser ML, Schoeller DA, Mossavar-Rahmani Y, Snetselaar LG, Van Horn LV, Eaton CB, Prentice RL, Lampe JW, O'Brien DM. The Carbon Isotope Ratios of Serum Amino Acids in Combination with Participant Characteristics can be Used to Estimate Added Sugar Intake in a Controlled Feeding Study of US Postmenopausal Women. J Nutr. 2020 Oct 12;150(10):2764-2771. doi: 10.1093/jn/nxaa195. PMID 32712658
- [Derived] Hooper L, Martin N, Jimoh OF, Kirk C, Foster E, Abdelhamid AS. Reduction in saturated fat intake for cardiovascular disease. Cochrane Database Syst Rev. 2020 May 19;5(5):CD011737. doi: 10.1002/14651858.CD011737.pub2. PMID 32428300
- [Derived] Manson JE, Bassuk SS, Kaunitz AM, Pinkerton JV. The Women's Health Initiative trials of menopausal hormone therapy: lessons learned. Menopause. 2020 Aug;27(8):918-928. doi: 10.1097/GME.0000000000001553. PMID 32345788
- [Derived] Van Horn L, Aragaki AK, Howard BV, Allison MA, Isasi CR, Manson JE, Neuhouser ML, Mossavar-Rahmani Y, Thomson CA, Vitolin MZ, Wallace RB, Prentice RL; WHI Investigators. Eating Pattern Response to a Low-Fat Diet Intervention and Cardiovascular Outcomes in Normotensive Women: The Women's Health Initiative. Curr Dev Nutr. 2020 Feb 12;4(3):nzaa021. doi: 10.1093/cdn/nzaa021. eCollection 2020 Mar. PMID 32159070
- [Derived] Chlebowski RT, Aragaki AK, Anderson GL, Pan K, Neuhouser ML, Manson JE, Thomson CA, Mossavar-Rahmani Y, Lane DS, Johnson KC, Wactawski-Wende J, Snetselaar L, Rohan TE, Luo J, Barac A, Prentice RL; Women's Health Initiative. Dietary Modification and Breast Cancer Mortality: Long-Term Follow-Up of the Women's Health Initiative Randomized Trial. J Clin Oncol. 2020 May 1;38(13):1419-1428. doi: 10.1200/JCO.19.00435. Epub 2020 Feb 7. PMID 32031879
- [Derived] Chlebowski RT, Rapp S, Aragaki AK, Pan K, Neuhouser ML, Snetselaar LG, Manson JE, Wactawski-Wende J, Johnson KC, Hayden K, Baker LD, Henderson VW, Garcia L, Qi L, Prentice RL. Low-fat dietary pattern and global cognitive function: Exploratory analyses of the Women's Health Initiative (WHI) randomized Dietary Modification trial. EClinicalMedicine. 2020 Jan 8;18:100240. doi: 10.1016/j.eclinm.2019.100240. eCollection 2020 Jan. PMID 31938786
- [Derived] Liu L, Klein L, Eaton C, Panjrath G, Martin LW, Chae CU, Greenland P, Lloyd-Jones DM, Wactawski-Wende J, Manson JE. Menopausal Hormone Therapy and Risks of First Hospitalized Heart Failure and its Subtypes During the Intervention and Extended Postintervention Follow-up of the Women's Health Initiative Randomized Trials. J Card Fail. 2020 Jan;26(1):2-12. doi: 10.1016/j.cardfail.2019.09.006. Epub 2019 Sep 17. PMID 31536806
- [Derived] Manson JE, Aragaki AK, Bassuk SS, Chlebowski RT, Anderson GL, Rossouw JE, Howard BV, Thomson CA, Stefanick ML, Kaunitz AM, Crandall CJ, Eaton CB, Henderson VW, Liu S, Luo J, Rohan T, Shadyab AH, Wells G, Wactawski-Wende J, Prentice RL; WHI Investigators. Menopausal Estrogen-Alone Therapy and Health Outcomes in Women With and Without Bilateral Oophorectomy: A Randomized Trial. Ann Intern Med. 2019 Sep 17;171(6):406-414. doi: 10.7326/M19-0274. Epub 2019 Sep 10. PMID 31499528
- [Derived] Prentice RL, Aragaki AK, Howard BV, Chlebowski RT, Thomson CA, Van Horn L, Tinker LF, Manson JE, Anderson GL, Kuller LE, Neuhouser ML, Johnson KC, Snetselaar L, Rossouw JE. Low-Fat Dietary Pattern among Postmenopausal Women Influences Long-Term Cancer, Cardiovascular Disease, and Diabetes Outcomes. J Nutr. 2019 Sep 1;149(9):1565-1574. doi: 10.1093/jn/nxz107. PMID 31175807
- [Derived] Jiang X, Nudy M, Aragaki AK, Robbins JA, Manson JE, Stefanick ML, O'Sullivan DM, Shikany JM, LeBlanc ES, Kelsey AM, Cauley J, Martin LW, Payne ME, Johnson KC, Howard B, Schnatz PF. Women's Health Initiative clinical trials: potential interactive effect of calcium and vitamin D supplementation with hormonal therapy on cardiovascular disease. Menopause. 2019 Aug;26(8):841-849. doi: 10.1097/GME.0000000000001360. PMID 31145202
- [Derived] Haring B, Crandall CJ, Carbone L, Liu S, Li W, Johnson KC, Wactawski-Wende J, Shadyab AH, Gass ML, Kamensky V, Cauley JA, Wassertheil-Smoller S. Lipoprotein(a) plasma levels, bone mineral density and risk of hip fracture: a post hoc analysis of the Women's Health Initiative, USA. BMJ Open. 2019 Apr 24;9(4):e027257. doi: 10.1136/bmjopen-2018-027257. PMID 31023762
- [Derived] Prentice RL, Pettinger M, Neuhouser ML, Tinker LF, Huang Y, Zheng C, Manson JE, Mossavar-Rahmani Y, Anderson GL, Lampe JW. Application of blood concentration biomarkers in nutritional epidemiology: example of carotenoid and tocopherol intake in relation to chronic disease risk. Am J Clin Nutr. 2019 Apr 1;109(4):1189-1196. doi: 10.1093/ajcn/nqy360. PMID 30915444
- [Derived] Felix AS, Lehman A, Nolan TS, Sealy-Jefferson S, Breathett K, Hood DB, Addison D, Anderson CM, Cene CW, Warren BJ, Jackson RD, Williams KP. Stress, Resilience, and Cardiovascular Disease Risk Among Black Women. Circ Cardiovasc Qual Outcomes. 2019 Apr;12(4):e005284. doi: 10.1161/CIRCOUTCOMES.118.005284. PMID 30909729
- [Derived] Prentice RL. Intake biomarkers and the chronic disease nutritional epidemiology research agenda. Am J Clin Nutr. 2018 Sep 1;108(3):433-434. doi: 10.1093/ajcn/nqy206. No abstract available. PMID 30535112
- [Derived] Iyengar NM, Arthur R, Manson JE, Chlebowski RT, Kroenke CH, Peterson L, Cheng TD, Feliciano EC, Lane D, Luo J, Nassir R, Pan K, Wassertheil-Smoller S, Kamensky V, Rohan TE, Dannenberg AJ. Association of Body Fat and Risk of Breast Cancer in Postmenopausal Women With Normal Body Mass Index: A Secondary Analysis of a Randomized Clinical Trial and Observational Study. JAMA Oncol. 2019 Feb 1;5(2):155-163. doi: 10.1001/jamaoncol.2018.5327. PMID 30520976
- [Derived] Al-Rousan T, Sparks JA, Pettinger M, Chlebowski R, Manson JE, Kauntiz AM, Wallace R. Menopausal hormone therapy and the incidence of carpal tunnel syndrome in postmenopausal women: Findings from the Women's Health Initiative. PLoS One. 2018 Dec 4;13(12):e0207509. doi: 10.1371/journal.pone.0207509. eCollection 2018. PMID 30513095
- [Derived] Yun HY, Lampe JW, Tinker LF, Neuhouser ML, Beresford SAA, Niles KR, Mossavar-Rahmani Y, Snetselaar LG, Van Horn L, Prentice RL, O'Brien DM. Serum Nitrogen and Carbon Stable Isotope Ratios Meet Biomarker Criteria for Fish and Animal Protein Intake in a Controlled Feeding Study of a Women's Health Initiative Cohort. J Nutr. 2018 Dec 1;148(12):1931-1937. doi: 10.1093/jn/nxy168. PMID 30239866
- [Derived] Parikh NI, Kapphahn K, Hedlin H, Olgin JE, Allison MA, Magnani JW, Ryckman KR, Waring ME, Perez MV, Howard BV. Effects of reproductive period duration and number of pregnancies on midlife ECG indices: a secondary analysis from the Women's Health Initiative Clinical Trial. BMJ Open. 2018 Aug 17;8(8):e019129. doi: 10.1136/bmjopen-2017-019129. PMID 30121588
- [Derived] Mora S, Wenger NK, Cook NR, Liu J, Howard BV, Limacher MC, Liu S, Margolis KL, Martin LW, Paynter NP, Ridker PM, Robinson JG, Rossouw JE, Safford MM, Manson JE. Evaluation of the Pooled Cohort Risk Equations for Cardiovascular Risk Prediction in a Multiethnic Cohort From the Women's Health Initiative. JAMA Intern Med. 2018 Sep 1;178(9):1231-1240. doi: 10.1001/jamainternmed.2018.2875. PMID 30039172
- [Derived] Chlebowski RT, Aragaki AK, Anderson GL, Simon MS, Manson JE, Neuhouser ML, Pan K, Stefanic ML, Rohan TE, Lane D, Qi L, Snetselaar L, Prentice RL. Association of Low-Fat Dietary Pattern With Breast Cancer Overall Survival: A Secondary Analysis of the Women's Health Initiative Randomized Clinical Trial. JAMA Oncol. 2018 Oct 1;4(10):e181212. doi: 10.1001/jamaoncol.2018.1212. Epub 2018 Oct 11. PMID 29800122
- [Derived] Shreibati JB, Manson JE, Margolis KL, Chlebowski RT, Stefanick ML, Hlatky MA. Impact of hormone therapy on Medicare spending in the Women's Health Initiative randomized clinical trials. Am Heart J. 2018 Apr;198:108-114. doi: 10.1016/j.ahj.2017.12.016. Epub 2017 Dec 27. PMID 29653631
- [Derived] Howard BV, Aragaki AK, Tinker LF, Allison M, Hingle MD, Johnson KC, Manson JE, Shadyab AH, Shikany JM, Snetselaar LG, Thomson CA, Zaslavsky O, Prentice RL. A Low-Fat Dietary Pattern and Diabetes: A Secondary Analysis From the Women's Health Initiative Dietary Modification Trial. Diabetes Care. 2018 Apr;41(4):680-687. doi: 10.2337/dc17-0534. Epub 2017 Dec 27. PMID 29282203
- [Derived] Gray KE, Katon JG, LeBlanc ES, Woods NF, Bastian LA, Reiber GE, Weitlauf JC, Nelson KM, LaCroix AZ. Vasomotor symptom characteristics: are they risk factors for incident diabetes? Menopause. 2018 May;25(5):520-530. doi: 10.1097/GME.0000000000001033. PMID 29206771
- [Derived] Poornima IG, Mackey RH, Allison MA, Manson JE, Carr JJ, LaMonte MJ, Chang Y, Kuller LH; WHI and WHI-CAC Study Investigators. Coronary Artery Calcification (CAC) and Post-Trial Cardiovascular Events and Mortality Within the Women's Health Initiative (WHI) Estrogen-Alone Trial. J Am Heart Assoc. 2017 Oct 27;6(11):e006887. doi: 10.1161/JAHA.117.006887. PMID 29079563
- [Derived] Jiao L, Chen L, White DL, Tinker L, Chlebowski RT, Van Horn LV, Richardson P, Lane D, Sangi-Haghpeykar H, El-Serag HB. Low-fat Dietary Pattern and Pancreatic Cancer Risk in the Women's Health Initiative Dietary Modification Randomized Controlled Trial. J Natl Cancer Inst. 2018 Jan 1;110(1):49-56. doi: 10.1093/jnci/djx117. PMID 28922784
- [Derived] Manson JE, Aragaki AK, Rossouw JE, Anderson GL, Prentice RL, LaCroix AZ, Chlebowski RT, Howard BV, Thomson CA, Margolis KL, Lewis CE, Stefanick ML, Jackson RD, Johnson KC, Martin LW, Shumaker SA, Espeland MA, Wactawski-Wende J; WHI Investigators. Menopausal Hormone Therapy and Long-term All-Cause and Cause-Specific Mortality: The Women's Health Initiative Randomized Trials. JAMA. 2017 Sep 12;318(10):927-938. doi: 10.1001/jama.2017.11217. PMID 28898378
- [Derived] Prentice RL, Aragaki AK, Van Horn L, Thomson CA, Beresford SA, Robinson J, Snetselaar L, Anderson GL, Manson JE, Allison MA, Rossouw JE, Howard BV. Low-fat dietary pattern and cardiovascular disease: results from the Women's Health Initiative randomized controlled trial. Am J Clin Nutr. 2017 Jul;106(1):35-43. doi: 10.3945/ajcn.117.153270. Epub 2017 May 17. PMID 28515068
- [Derived] Song X, Huang Y, Neuhouser ML, Tinker LF, Vitolins MZ, Prentice RL, Lampe JW. Dietary long-chain fatty acids and carbohydrate biomarker evaluation in a controlled feeding study in participants from the Women's Health Initiative cohort. Am J Clin Nutr. 2017 Jun;105(6):1272-1282. doi: 10.3945/ajcn.117.153072. Epub 2017 Apr 26. PMID 28446501
- [Derived] Harris WS, Luo J, Pottala JV, Espeland MA, Margolis KL, Manson JE, Wang L, Brasky TM, Robinson JG. Red blood cell polyunsaturated fatty acids and mortality in the Women's Health Initiative Memory Study. J Clin Lipidol. 2017 Jan-Feb;11(1):250-259.e5. doi: 10.1016/j.jacl.2016.12.013. Epub 2017 Jan 12. PMID 28391893
- [Derived] Gourlay ML, Overman RA, Fine JP, Crandall CJ, Robbins J, Schousboe JT, Ensrud KE, LeBlanc ES, Gass ML, Johnson KC, Womack CR, LaCroix AZ; Women's Health Initiative Investigators. Time to Clinically Relevant Fracture Risk Scores in Postmenopausal Women. Am J Med. 2017 Jul;130(7):862.e15-862.e23. doi: 10.1016/j.amjmed.2017.02.012. Epub 2017 Mar 9. PMID 28285070
- [Derived] LaCroix AZ, Rillamas-Sun E, Buchner D, Evenson KR, Di C, Lee IM, Marshall S, LaMonte MJ, Hunt J, Tinker LF, Stefanick M, Lewis CE, Bellettiere J, Herring AH. The Objective Physical Activity and Cardiovascular Disease Health in Older Women (OPACH) Study. BMC Public Health. 2017 Feb 14;17(1):192. doi: 10.1186/s12889-017-4065-6. PMID 28193194
- [Derived] Lampe JW, Huang Y, Neuhouser ML, Tinker LF, Song X, Schoeller DA, Kim S, Raftery D, Di C, Zheng C, Schwarz Y, Van Horn L, Thomson CA, Mossavar-Rahmani Y, Beresford SA, Prentice RL. Dietary biomarker evaluation in a controlled feeding study in women from the Women's Health Initiative cohort. Am J Clin Nutr. 2017 Feb;105(2):466-475. doi: 10.3945/ajcn.116.144840. Epub 2016 Dec 28. PMID 28031191
- [Derived] Schnatz PF, Jiang X, Aragaki AK, Nudy M, O'Sullivan DM, Williams M, LeBlanc ES, Martin LW, Manson JE, Shikany JM, Johnson KC, Stefanick ML, Payne ME, Cauley JA, Howard BV, Robbins J. Effects of Calcium, Vitamin D, and Hormone Therapy on Cardiovascular Disease Risk Factors in the Women's Health Initiative: A Randomized Controlled Trial. Obstet Gynecol. 2017 Jan;129(1):121-129. doi: 10.1097/AOG.0000000000001774. PMID 27926633
- [Derived] Chlebowski RT, Barrington W, Aragaki AK, Manson JE, Sarto G, O'Sullivan MJ, Wu D, Cauley JA, Qi L, Wallace RL, Prentice RL. Estrogen alone and health outcomes in black women by African ancestry: a secondary analyses of a randomized controlled trial. Menopause. 2017 Feb;24(2):133-141. doi: 10.1097/GME.0000000000000733. PMID 27749739
- [Derived] Eaton CB, Pettinger M, Rossouw J, Martin LW, Foraker R, Quddus A, Liu S, Wampler NS, Hank Wu WC, Manson JE, Margolis K, Johnson KC, Allison M, Corbie-Smith G, Rosamond W, Breathett K, Klein L. Risk Factors for Incident Hospitalized Heart Failure With Preserved Versus Reduced Ejection Fraction in a Multiracial Cohort of Postmenopausal Women. Circ Heart Fail. 2016 Oct;9(10):e002883. doi: 10.1161/CIRCHEARTFAILURE.115.002883. PMID 27682440
- [Derived] Garcia DO, Lander EM, Wertheim BC, Manson JE, Volpe SL, Chlebowski RT, Stefanick ML, Lessin LS, Kuller LH, Thomson CA. Pet Ownership and Cancer Risk in the Women's Health Initiative. Cancer Epidemiol Biomarkers Prev. 2016 Sep;25(9):1311-6. doi: 10.1158/1055-9965.EPI-16-0218. Epub 2016 Jun 30. PMID 27365150
- [Derived] Zambrana RE, Lopez L, Dinwiddie GY, Ray RM, Eaton CB, Phillips LS, Wassertheil-Smoller S. Association of Baseline Depressive Symptoms with Prevalent and Incident Pre-Hypertension and Hypertension in Postmenopausal Hispanic Women: Results from the Women's Health Initiative. PLoS One. 2016 Apr 28;11(4):e0152765. doi: 10.1371/journal.pone.0152765. eCollection 2016. PMID 27124184
- [Derived] Wang A, Stefanick ML, Kapphahn K, Hedlin H, Desai M, Manson JA, Strickler H, Martin L, Wactawski-Wende J, Simon M, Tang JY. Relation of statin use with non-melanoma skin cancer: prospective results from the Women's Health Initiative. Br J Cancer. 2016 Feb 2;114(3):314-20. doi: 10.1038/bjc.2015.376. Epub 2016 Jan 7. PMID 26742009
- [Derived] Allison MA, Aragaki AK, Ray RM, Margolis KL, Beresford SA, Kuller L, Jo O'Sullivan M, Wassertheil-Smoller S, Van Horn L. A Randomized Trial of a Low-Fat Diet Intervention on Blood Pressure and Hypertension: Tertiary Analysis of the WHI Dietary Modification Trial. Am J Hypertens. 2016 Aug;29(8):959-68. doi: 10.1093/ajh/hpv196. Epub 2015 Dec 26. PMID 26708006
- [Derived] Johnson KC, Aragaki AK, Jackson R, Reiner A, Sandset PM, Rosing J, Dahm AE, Rosendaal F, Manson JE, Martin LW, Liu S, Kuller LH, Cushman M, Rossouw JE. Tissue Factor Pathway Inhibitor, Activated Protein C Resistance, and Risk of Coronary Heart Disease Due To Combined Estrogen Plus Progestin Therapy. Arterioscler Thromb Vasc Biol. 2016 Feb;36(2):418-24. doi: 10.1161/ATVBAHA.115.306905. Epub 2015 Dec 17. PMID 26681757
- [Derived] Espeland MA, Brinton RD, Hugenschmidt C, Manson JE, Craft S, Yaffe K, Weitlauf J, Vaughan L, Johnson KC, Padula CB, Jackson RD, Resnick SM; WHIMS Study Group. Impact of Type 2 Diabetes and Postmenopausal Hormone Therapy on Incidence of Cognitive Impairment in Older Women. Diabetes Care. 2015 Dec;38(12):2316-24. doi: 10.2337/dc15-1385. Epub 2015 Oct 20. PMID 26486190
- [Derived] Assaf AR, Beresford SAA, Risica PM, Aragaki A, Brunner RL, Bowen DJ, Naughton M, Rosal MC, Snetselaar L, Wenger N. Low-Fat Dietary Pattern Intervention and Health-Related Quality of Life: The Women's Health Initiative Randomized Controlled Dietary Modification Trial. J Acad Nutr Diet. 2016 Feb;116(2):259-271. doi: 10.1016/j.jand.2015.07.016. Epub 2015 Sep 16. PMID 26384466
- [Derived] Neuhouser ML, Aragaki AK, Prentice RL, Manson JE, Chlebowski R, Carty CL, Ochs-Balcom HM, Thomson CA, Caan BJ, Tinker LF, Urrutia RP, Knudtson J, Anderson GL. Overweight, Obesity, and Postmenopausal Invasive Breast Cancer Risk: A Secondary Analysis of the Women's Health Initiative Randomized Clinical Trials. JAMA Oncol. 2015 Aug;1(5):611-21. doi: 10.1001/jamaoncol.2015.1546. PMID 26182172
- [Derived] Ing SW, Orchard TS, Lu B, LaMonte MJ, Barbour KE, Cauley JA, Jackson RD. TNF Receptors Predict Hip Fracture Risk in the WHI Study and Fatty Acid Intake Does Not Modify This Association. J Clin Endocrinol Metab. 2015 Sep;100(9):3380-7. doi: 10.1210/JC.2015-1662. Epub 2015 Jul 10. PMID 26161450
- [Derived] Rillamas-Sun E, Buchner DM, Di C, Evenson KR, LaCroix AZ. Development and application of an automated algorithm to identify a window of consecutive days of accelerometer wear for large-scale studies. BMC Res Notes. 2015 Jun 26;8:270. doi: 10.1186/s13104-015-1229-2. PMID 26113170
- [Derived] Gangwisch JE, Hale L, Garcia L, Malaspina D, Opler MG, Payne ME, Rossom RC, Lane D. High glycemic index diet as a risk factor for depression: analyses from the Women's Health Initiative. Am J Clin Nutr. 2015 Aug;102(2):454-63. doi: 10.3945/ajcn.114.103846. Epub 2015 Jun 24. PMID 26109579
- [Derived] Schmiegelow MD, Hedlin H, Stefanick ML, Mackey RH, Allison M, Martin LW, Robinson JG, Hlatky MA. Insulin Resistance and Risk of Cardiovascular Disease in Postmenopausal Women: A Cohort Study From the Women's Health Initiative. Circ Cardiovasc Qual Outcomes. 2015 May;8(3):309-16. doi: 10.1161/CIRCOUTCOMES.114.001563. Epub 2015 May 5. PMID 25944628
- [Derived] Brasky TM, Rodabough RJ, Liu J, Kurta ML, Wise LA, Orchard TS, Cohn DE, Belury MA, White E, Manson JE, Neuhouser ML. Long-chain omega-3 fatty acid intake and endometrial cancer risk in the Women's Health Initiative. Am J Clin Nutr. 2015 Apr;101(4):824-34. doi: 10.3945/ajcn.114.098988. Epub 2015 Mar 4. PMID 25739930
- [Derived] Zubair N, Kooperberg C, Liu J, Di C, Peters U, Neuhouser ML. Genetic variation predicts serum lycopene concentrations in a multiethnic population of postmenopausal women. J Nutr. 2015 Feb;145(2):187-92. doi: 10.3945/jn.114.202150. Epub 2014 Dec 3. PMID 25644336
- [Derived] Donneyong MM, Hornung CA, Taylor KC, Baumgartner RN, Myers JA, Eaton CB, Gorodeski EZ, Klein L, Martin LW, Shikany JM, Song Y, Li W, Manson JE. Risk of heart failure among postmenopausal women: a secondary analysis of the randomized trial of vitamin D plus calcium of the women's health initiative. Circ Heart Fail. 2015 Jan;8(1):49-56. doi: 10.1161/CIRCHEARTFAILURE.114.001738. Epub 2014 Nov 14. PMID 25398967
- [Derived] Gourlay ML, Overman RA, Fine JP, Ensrud KE, Crandall CJ, Gass ML, Robbins J, Johnson KC, LeBlanc ES, Womack CR, Schousboe JT, LaCroix AZ; Women's Health Initiative Investigators. Baseline age and time to major fracture in younger postmenopausal women. Menopause. 2015 Jun;22(6):589-97. doi: 10.1097/GME.0000000000000356. PMID 25349960
- [Derived] Wang A, Kubo J, Luo J, Desai M, Hedlin H, Henderson M, Chlebowski R, Tindle H, Chen C, Gomez S, Manson JE, Schwartz AG, Wactawski-Wende J, Cote M, Patel MI, Stefanick ML, Wakelee HA. Active and passive smoking in relation to lung cancer incidence in the Women's Health Initiative Observational Study prospective cohort. Ann Oncol. 2015 Jan;26(1):221-230. doi: 10.1093/annonc/mdu470. Epub 2014 Oct 14. PMID 25316260
- [Derived] Rautaharju PM, Zhang ZM, Vitolins M, Perez M, Allison MA, Greenland P, Soliman EZ. Electrocardiographic repolarization-related variables as predictors of coronary heart disease death in the women's health initiative study. J Am Heart Assoc. 2014 Jul 28;3(4):e001005. doi: 10.1161/JAHA.114.001005. PMID 25074699
- [Derived] Bavry AA, Thomas F, Allison M, Johnson KC, Howard BV, Hlatky M, Manson JE, Limacher MC. Nonsteroidal anti-inflammatory drugs and cardiovascular outcomes in women: results from the women's health initiative. Circ Cardiovasc Qual Outcomes. 2014 Jul;7(4):603-10. doi: 10.1161/CIRCOUTCOMES.113.000800. Epub 2014 Jul 8. PMID 25006185
- [Derived] Shimbo D, Wang L, Lamonte MJ, Allison M, Wellenius GA, Bavry AA, Martin LW, Aragaki A, Newman JD, Swica Y, Rossouw JE, Manson JE, Wassertheil-Smoller S. The effect of hormone therapy on mean blood pressure and visit-to-visit blood pressure variability in postmenopausal women: results from the Women's Health Initiative randomized controlled trials. J Hypertens. 2014 Oct;32(10):2071-81; discussion 2081. doi: 10.1097/HJH.0000000000000287. PMID 24991872
- [Derived] Kabat GC, Heo M, Allison MA, Hou L, Nassir R, Zaslavsky O, Rohan TE. Association of anthropometric measures and hemostatic factors in postmenopausal women: a longitudinal study. Nutr Metab Cardiovasc Dis. 2014 Oct;24(10):1120-7. doi: 10.1016/j.numecd.2014.04.008. Epub 2014 May 2. PMID 24880739
- [Derived] Allison MA, Aragaki A, Eaton C, Li W, Van Horn L, Daviglus ML, Berger JS. Effect of dietary modification on incident carotid artery disease in postmenopausal women: results from the women's health initiative dietary modification trial. Stroke. 2014 Jun;45(6):1748-56. doi: 10.1161/STROKEAHA.114.005096. Epub 2014 Apr 17. PMID 24743440
- [Derived] Zhao S, Chlebowski RT, Anderson GL, Kuller LH, Manson JE, Gass M, Patterson R, Rohan TE, Lane DS, Beresford SA, Lavasani S, Rossouw JE, Prentice RL. Sex hormone associations with breast cancer risk and the mediation of randomized trial postmenopausal hormone therapy effects. Breast Cancer Res. 2014 Mar 26;16(2):R30. doi: 10.1186/bcr3632. PMID 24670297
- [Derived] Abbenhardt C, Miller JW, Song X, Brown EC, Cheng TY, Wener MH, Zheng Y, Toriola AT, Neuhouser ML, Beresford SA, Makar KW, Bailey LB, Maneval DR, Green R, Manson JE, Van Horn L, Ulrich CM. Biomarkers of one-carbon metabolism are associated with biomarkers of inflammation in women. J Nutr. 2014 May;144(5):714-21. doi: 10.3945/jn.113.183970. Epub 2014 Mar 19. PMID 24647390
- [Derived] Beasley JM, LaCroix AZ, Larson JC, Huang Y, Neuhouser ML, Tinker LF, Jackson R, Snetselaar L, Johnson KC, Eaton CB, Prentice RL. Biomarker-calibrated protein intake and bone health in the Women's Health Initiative clinical trials and observational study. Am J Clin Nutr. 2014 Apr;99(4):934-40. doi: 10.3945/ajcn.113.076786. Epub 2014 Feb 19. PMID 24552750
- [Derived] Orchard TS, Larson JC, Alghothani N, Bout-Tabaku S, Cauley JA, Chen Z, LaCroix AZ, Wactawski-Wende J, Jackson RD. Magnesium intake, bone mineral density, and fractures: results from the Women's Health Initiative Observational Study. Am J Clin Nutr. 2014 Apr;99(4):926-33. doi: 10.3945/ajcn.113.067488. Epub 2014 Feb 5. PMID 24500155
- [Derived] Zambrana RE, Lopez L, Dinwiddie GY, Ray RM, Phillips LS, Trevisan M, Wassertheil-Smoller S. Prevalence and incident prehypertension and hypertension in postmenopausal Hispanic women: results from the Women's Health Initiative. Am J Hypertens. 2014 Mar;27(3):372-81. doi: 10.1093/ajh/hpt279. Epub 2014 Jan 30. PMID 24480867
- [Derived] Hlatky MA, Ray RM, Burwen DR, Margolis KL, Johnson KC, Kucharska-Newton A, Manson JE, Robinson JG, Safford MM, Allison M, Assimes TL, Bavry AA, Berger J, Cooper-DeHoff RM, Heckbert SR, Li W, Liu S, Martin LW, Perez MV, Tindle HA, Winkelmayer WC, Stefanick ML. Use of Medicare data to identify coronary heart disease outcomes in the Women's Health Initiative. Circ Cardiovasc Qual Outcomes. 2014 Jan;7(1):157-62. doi: 10.1161/CIRCOUTCOMES.113.000373. Epub 2014 Jan 7. PMID 24399330
- [Derived] Prentice RL, Zhao S, Johnson M, Aragaki A, Hsia J, Jackson RD, Rossouw JE, Manson JE, Hanash SM. Proteomic risk markers for coronary heart disease and stroke: validation and mediation of randomized trial hormone therapy effects on these diseases. Genome Med. 2013 Dec 27;5(12):112. doi: 10.1186/gm517. eCollection 2013. PMID 24373343
- [Derived] Bertoia ML, Triche EW, Michaud DS, Baylin A, Hogan JW, Neuhouser ML, Tinker LF, Van Horn L, Waring ME, Li W, Shikany JM, Eaton CB. Mediterranean and Dietary Approaches to Stop Hypertension dietary patterns and risk of sudden cardiac death in postmenopausal women. Am J Clin Nutr. 2014 Feb;99(2):344-51. doi: 10.3945/ajcn.112.056135. Epub 2013 Dec 18. PMID 24351877
- [Derived] Huang Y, Van Horn L, Tinker LF, Neuhouser ML, Carbone L, Mossavar-Rahmani Y, Thomas F, Prentice RL. Measurement error corrected sodium and potassium intake estimation using 24-hour urinary excretion. Hypertension. 2014 Feb;63(2):238-44. doi: 10.1161/HYPERTENSIONAHA.113.02218. Epub 2013 Nov 25. PMID 24277763
- [Derived] Levitan EB, Lewis CE, Tinker LF, Eaton CB, Ahmed A, Manson JE, Snetselaar LG, Martin LW, Trevisan M, Howard BV, Shikany JM. Mediterranean and DASH diet scores and mortality in women with heart failure: The Women's Health Initiative. Circ Heart Fail. 2013 Nov;6(6):1116-23. doi: 10.1161/CIRCHEARTFAILURE.113.000495. Epub 2013 Oct 9. PMID 24107587
- [Derived] Manson JE, Chlebowski RT, Stefanick ML, Aragaki AK, Rossouw JE, Prentice RL, Anderson G, Howard BV, Thomson CA, LaCroix AZ, Wactawski-Wende J, Jackson RD, Limacher M, Margolis KL, Wassertheil-Smoller S, Beresford SA, Cauley JA, Eaton CB, Gass M, Hsia J, Johnson KC, Kooperberg C, Kuller LH, Lewis CE, Liu S, Martin LW, Ockene JK, O'Sullivan MJ, Powell LH, Simon MS, Van Horn L, Vitolins MZ, Wallace RB. Menopausal hormone therapy and health outcomes during the intervention and extended poststopping phases of the Women's Health Initiative randomized trials. JAMA. 2013 Oct 2;310(13):1353-68. doi: 10.1001/jama.2013.278040. PMID 24084921
- [Derived] Cheng TY, Lacroix AZ, Beresford SA, Goodman GE, Thornquist MD, Zheng Y, Chlebowski RT, Ho GY, Neuhouser ML. Vitamin D intake and lung cancer risk in the Women's Health Initiative. Am J Clin Nutr. 2013 Oct;98(4):1002-11. doi: 10.3945/ajcn.112.055905. Epub 2013 Aug 21. PMID 23966428
- [Derived] Zhang ZM, Rautaharju PM, Soliman EZ, Manson JE, Martin LW, Perez M, Vitolins M, Prineas RJ. Different patterns of bundle-branch blocks and the risk of incident heart failure in the Women's Health Initiative (WHI) study. Circ Heart Fail. 2013 Jul;6(4):655-61. doi: 10.1161/CIRCHEARTFAILURE.113.000217. Epub 2013 May 31. PMID 23729198
- [Derived] Gamba CS, Stefanick ML, Shikany JM, Larson J, Linos E, Sims ST, Marshall J, Van Horn L, Zeitouni N, Tang JY. Low-fat diet and skin cancer risk: the women's health initiative randomized controlled dietary modification trial. Cancer Epidemiol Biomarkers Prev. 2013 Sep;22(9):1509-19. doi: 10.1158/1055-9965.EPI-13-0341. Epub 2013 May 22. PMID 23697610
- [Derived] Mossavar-Rahmani Y, Tinker LF, Huang Y, Neuhouser ML, McCann SE, Seguin RA, Vitolins MZ, Curb JD, Prentice RL. Factors relating to eating style, social desirability, body image and eating meals at home increase the precision of calibration equations correcting self-report measures of diet using recovery biomarkers: findings from the Women's Health Initiative. Nutr J. 2013 May 16;12:63. doi: 10.1186/1475-2891-12-63. PMID 23679960
- [Derived] Bertoia ML, Triche EW, Michaud DS, Baylin A, Hogan JW, Neuhouser ML, Freiberg MS, Allison MA, Safford MM, Li W, Mossavar-Rahmani Y, Rosal MC, Eaton CB. Long-term alcohol and caffeine intake and risk of sudden cardiac death in women. Am J Clin Nutr. 2013 Jun;97(6):1356-63. doi: 10.3945/ajcn.112.044248. Epub 2013 Apr 24. PMID 23615825
- [Derived] Gamba CA, Swetter SM, Stefanick ML, Kubo J, Desai M, Spaunhurst KM, Sinha AA, Asgari MM, Sturgeon S, Tang JY. Aspirin is associated with lower melanoma risk among postmenopausal Caucasian women: the Women's Health Initiative. Cancer. 2013 Apr 15;119(8):1562-9. doi: 10.1002/cncr.27817. Epub 2013 Mar 11. PMID 23483536
- [Derived] Espeland MA, Pettinger M, Falkner KL, Shumaker SA, Limacher M, Thomas F, Weaver KE, Stefanick ML, McQuellon C, Hunt JR, Johnson KC. Demographic and health factors associated with enrollment in posttrial studies: the Women's Health Initiative Hormone Therapy Trials. Clin Trials. 2013;10(3):463-72. doi: 10.1177/1740774513477931. Epub 2013 Mar 12. PMID 23480899
- [Derived] Miller JW, Beresford SA, Neuhouser ML, Cheng TY, Song X, Brown EC, Zheng Y, Rodriguez B, Green R, Ulrich CM. Homocysteine, cysteine, and risk of incident colorectal cancer in the Women's Health Initiative observational cohort. Am J Clin Nutr. 2013 Apr;97(4):827-34. doi: 10.3945/ajcn.112.049932. Epub 2013 Feb 20. PMID 23426034
- [Derived] Fesinmeyer MD, North KE, Lim U, Buzkova P, Crawford DC, Haessler J, Gross MD, Fowke JH, Goodloe R, Love SA, Graff M, Carlson CS, Kuller LH, Matise TC, Hong CP, Henderson BE, Allen M, Rohde RR, Mayo P, Schnetz-Boutaud N, Monroe KR, Ritchie MD, Prentice RL, Kolonel LN, Manson JE, Pankow J, Hindorff LA, Franceschini N, Wilkens LR, Haiman CA, Le Marchand L, Peters U. Effects of smoking on the genetic risk of obesity: the population architecture using genomics and epidemiology study. BMC Med Genet. 2013 Jan 11;14:6. doi: 10.1186/1471-2350-14-6. PMID 23311614
- [Derived] Perez MV, Wang PJ, Larson JC, Virnig BA, Cochrane B, Curb JD, Klein L, Manson JE, Martin LW, Robinson J, Wassertheil-Smoller S, Stefanick ML. Effects of postmenopausal hormone therapy on incident atrial fibrillation: the Women's Health Initiative randomized controlled trials. Circ Arrhythm Electrophysiol. 2012 Dec;5(6):1108-16. doi: 10.1161/CIRCEP.112.972224. Epub 2012 Nov 20. PMID 23169946
- [Derived] Orchard TS, Ing SW, Lu B, Belury MA, Johnson K, Wactawski-Wende J, Jackson RD. The association of red blood cell n-3 and n-6 fatty acids with bone mineral density and hip fracture risk in the women's health initiative. J Bone Miner Res. 2013 Mar;28(3):505-15. doi: 10.1002/jbmr.1772. PMID 23018646
- [Derived] Rossouw JE, Prentice RL, Manson JE, Aragaki AK, Hsia J, Martin LW, Kuller L, Johnson KC, Eaton C, Jackson R, Trevisan M, Allison M, Hoogeveen RC. Relationships of coronary heart disease with 27-hydroxycholesterol, low-density lipoprotein cholesterol, and menopausal hormone therapy. Circulation. 2012 Sep 25;126(13):1577-86. doi: 10.1161/CIRCULATIONAHA.112.103218. Epub 2012 Aug 29. PMID 22932256
- [Derived] Eaton CB, Abdulbaki AM, Margolis KL, Manson JE, Limacher M, Klein L, Allison MA, Robinson JG, Curb JD, Martin LA, Liu S, Howard BV. Racial and ethnic differences in incident hospitalized heart failure in postmenopausal women: the Women's Health Initiative. Circulation. 2012 Aug 7;126(6):688-96. doi: 10.1161/CIRCULATIONAHA.111.066688. Epub 2012 Jul 2. PMID 22753306
- [Derived] Interleukin-6 Receptor Mendelian Randomisation Analysis (IL6R MR) Consortium; Swerdlow DI, Holmes MV, Kuchenbaecker KB, Engmann JE, Shah T, Sofat R, Guo Y, Chung C, Peasey A, Pfister R, Mooijaart SP, Ireland HA, Leusink M, Langenberg C, Li KW, Palmen J, Howard P, Cooper JA, Drenos F, Hardy J, Nalls MA, Li YR, Lowe G, Stewart M, Bielinski SJ, Peto J, Timpson NJ, Gallacher J, Dunlop M, Houlston R, Tomlinson I, Tzoulaki I, Luan J, Boer JM, Forouhi NG, Onland-Moret NC, van der Schouw YT, Schnabel RB, Hubacek JA, Kubinova R, Baceviciene M, Tamosiunas A, Pajak A, Topor-Madry R, Malyutina S, Baldassarre D, Sennblad B, Tremoli E, de Faire U, Ferrucci L, Bandenelli S, Tanaka T, Meschia JF, Singleton A, Navis G, Mateo Leach I, Bakker SJ, Gansevoort RT, Ford I, Epstein SE, Burnett MS, Devaney JM, Jukema JW, Westendorp RG, Jan de Borst G, van der Graaf Y, de Jong PA, Mailand-van der Zee AH, Klungel OH, de Boer A, Doevendans PA, Stephens JW, Eaton CB, Robinson JG, Manson JE, Fowkes FG, Frayling TM, Price JF, Whincup PH, Morris RW, Lawlor DA, Smith GD, Ben-Shlomo Y, Redline S, Lange LA, Kumari M, Wareham NJ, Verschuren WM, Benjamin EJ, Whittaker JC, Hamsten A, Dudbridge F, Delaney JA, Wong A, Kuh D, Hardy R, Castillo BA, Connolly JJ, van der Harst P, Brunner EJ, Marmot MG, Wassel CL, Humphries SE, Talmud PJ, Kivimaki M, Asselbergs FW, Voevoda M, Bobak M, Pikhart H, Wilson JG, Hakonarson H, Reiner AP, Keating BJ, Sattar N, Hingorani AD, Casas JP. The interleukin-6 receptor as a target for prevention of coronary heart disease: a mendelian randomisation analysis. Lancet. 2012 Mar 31;379(9822):1214-24. doi: 10.1016/S0140-6736(12)60110-X. Epub 2012 Mar 14. PMID 22421340
- [Derived] Anderson GL, Chlebowski RT, Aragaki AK, Kuller LH, Manson JE, Gass M, Bluhm E, Connelly S, Hubbell FA, Lane D, Martin L, Ockene J, Rohan T, Schenken R, Wactawski-Wende J. Conjugated equine oestrogen and breast cancer incidence and mortality in postmenopausal women with hysterectomy: extended follow-up of the Women's Health Initiative randomised placebo-controlled trial. Lancet Oncol. 2012 May;13(5):476-86. doi: 10.1016/S1470-2045(12)70075-X. Epub 2012 Mar 7. PMID 22401913
- [Derived] Rossouw JE, Johnson KC, Pettinger M, Cushman M, Sandset PM, Kuller L, Rosendaal F, Rosing J, Wasserthal-Smoller S, Martin LW, Manson JE, Lakshminarayan K, Merino JG, Lynch J. Tissue factor pathway inhibitor, activated protein C resistance, and risk of ischemic stroke due to postmenopausal hormone therapy. Stroke. 2012 Apr;43(4):952-7. doi: 10.1161/STROKEAHA.111.643072. Epub 2012 Feb 23. PMID 22363056
- [Derived] Tinker LF, Sarto GE, Howard BV, Huang Y, Neuhouser ML, Mossavar-Rahmani Y, Beasley JM, Margolis KL, Eaton CB, Phillips LS, Prentice RL. Biomarker-calibrated dietary energy and protein intake associations with diabetes risk among postmenopausal women from the Women's Health Initiative. Am J Clin Nutr. 2011 Dec;94(6):1600-6. doi: 10.3945/ajcn.111.018648. Epub 2011 Nov 9. PMID 22071707
- [Derived] Eaton CB, Young A, Allison MA, Robinson J, Martin LW, Kuller LH, Johnson KC, Curb JD, Van Horn L, McTiernan A, Liu S, Manson JE. Prospective association of vitamin D concentrations with mortality in postmenopausal women: results from the Women's Health Initiative (WHI). Am J Clin Nutr. 2011 Dec;94(6):1471-8. doi: 10.3945/ajcn.111.017715. Epub 2011 Oct 26. PMID 22030222
- [Derived] Bolland MJ, Grey A, Gamble GD, Reid IR. Calcium and vitamin D supplements and health outcomes: a reanalysis of the Women's Health Initiative (WHI) limited-access data set. Am J Clin Nutr. 2011 Oct;94(4):1144-9. doi: 10.3945/ajcn.111.015032. Epub 2011 Aug 31. PMID 21880848
- [Derived] Prentice RL, Mossavar-Rahmani Y, Huang Y, Van Horn L, Beresford SA, Caan B, Tinker L, Schoeller D, Bingham S, Eaton CB, Thomson C, Johnson KC, Ockene J, Sarto G, Heiss G, Neuhouser ML. Evaluation and comparison of food records, recalls, and frequencies for energy and protein assessment by using recovery biomarkers. Am J Epidemiol. 2011 Sep 1;174(5):591-603. doi: 10.1093/aje/kwr140. Epub 2011 Jul 15. PMID 21765003
- [Derived] Eaton CB, Hochberg MC, Assaf A, Cryer BL, Lu B, Sands G, Rodriguez B, LaCroix A, Lessin L, Limacher MC, Fugate Woods N, Connelly S, Chen Z. The cross-sectional relationship of hemoglobin levels and functional outcomes in women with self-reported osteoarthritis: results from the Women's Health Initiative. Semin Arthritis Rheum. 2011 Dec;41(3):406-14. doi: 10.1016/j.semarthrit.2011.04.008. Epub 2011 Jul 2. PMID 21723591
- [Derived] Olsen CM, Pandeya N, Green AC, Webb PM, Whiteman DC; Australian Cancer Study. Population attributable fractions of adenocarcinoma of the esophagus and gastroesophageal junction. Am J Epidemiol. 2011 Sep 1;174(5):582-90. doi: 10.1093/aje/kwr117. Epub 2011 Jun 30. PMID 21719746
- [Derived] Harrow BS, Eaton CB, Roberts MB, Assaf AR, Luo X, Chen Z. Health utilities associated with hemoglobin levels and blood loss in postmenopausal women: the Women's Health Initiative. Value Health. 2011 Jun;14(4):555-63. doi: 10.1016/j.jval.2010.11.008. Epub 2011 Apr 30. PMID 21669380
- [Derived] Chacko SA, Song Y, Manson JE, Van Horn L, Eaton C, Martin LW, McTiernan A, Curb JD, Wylie-Rosett J, Phillips LS, Plodkowski RA, Liu S. Serum 25-hydroxyvitamin D concentrations in relation to cardiometabolic risk factors and metabolic syndrome in postmenopausal women. Am J Clin Nutr. 2011 Jul;94(1):209-17. doi: 10.3945/ajcn.110.010272. Epub 2011 May 25. PMID 21613558
- [Derived] Shikany JM, Margolis KL, Pettinger M, Jackson RD, Limacher MC, Liu S, Phillips LS, Tinker LF. Effects of a low-fat dietary intervention on glucose, insulin, and insulin resistance in the Women's Health Initiative (WHI) Dietary Modification trial. Am J Clin Nutr. 2011 Jul;94(1):75-85. doi: 10.3945/ajcn.110.010843. Epub 2011 May 11. PMID 21562091
- [Derived] Wallace RB, Wactawski-Wende J, O'Sullivan MJ, Larson JC, Cochrane B, Gass M, Masaki K. Urinary tract stone occurrence in the Women's Health Initiative (WHI) randomized clinical trial of calcium and vitamin D supplements. Am J Clin Nutr. 2011 Jul;94(1):270-7. doi: 10.3945/ajcn.110.003350. Epub 2011 Apr 27. PMID 21525191
- [Derived] LaCroix AZ, Chlebowski RT, Manson JE, Aragaki AK, Johnson KC, Martin L, Margolis KL, Stefanick ML, Brzyski R, Curb JD, Howard BV, Lewis CE, Wactawski-Wende J; WHI Investigators. Health outcomes after stopping conjugated equine estrogens among postmenopausal women with prior hysterectomy: a randomized controlled trial. JAMA. 2011 Apr 6;305(13):1305-14. doi: 10.1001/jama.2011.382. PMID 21467283
- [Derived] Gaussoin SA, Espeland MA, Absher J, Howard BV, Jones BM, Rapp SR. Ascertaining dementia-related outcomes for deceased or proxy-dependent participants: an overview of the Women's Health Initiative Memory Study supplemental case ascertainment protocol. Int J Geriatr Psychiatry. 2012 Feb;27(2):205-14. doi: 10.1002/gps.2714. Epub 2011 Mar 18. PMID 21416508
- [Derived] Carty CL, Kooperberg C, Neuhouser ML, Tinker L, Howard B, Wactawski-Wende J, Beresford SA, Snetselaar L, Vitolins M, Allison M, Budrys N, Prentice R, Peters U. Low-fat dietary pattern and change in body-composition traits in the Women's Health Initiative Dietary Modification Trial. Am J Clin Nutr. 2011 Mar;93(3):516-24. doi: 10.3945/ajcn.110.006395. Epub 2010 Dec 22. PMID 21177798
- [Derived] Orchard TS, Cauley JA, Frank GC, Neuhouser ML, Robinson JG, Snetselaar L, Tylavsky F, Wactawski-Wende J, Young AM, Lu B, Jackson RD. Fatty acid consumption and risk of fracture in the Women's Health Initiative. Am J Clin Nutr. 2010 Dec;92(6):1452-60. doi: 10.3945/ajcn.2010.29955. Epub 2010 Oct 27. PMID 20980487
- [Derived] Chlebowski RT, Anderson GL, Gass M, Lane DS, Aragaki AK, Kuller LH, Manson JE, Stefanick ML, Ockene J, Sarto GE, Johnson KC, Wactawski-Wende J, Ravdin PM, Schenken R, Hendrix SL, Rajkovic A, Rohan TE, Yasmeen S, Prentice RL; WHI Investigators. Estrogen plus progestin and breast cancer incidence and mortality in postmenopausal women. JAMA. 2010 Oct 20;304(15):1684-92. doi: 10.1001/jama.2010.1500. PMID 20959578
- [Derived] Maalouf NM, Sato AH, Welch BJ, Howard BV, Cochrane BB, Sakhaee K, Robbins JA. Postmenopausal hormone use and the risk of nephrolithiasis: results from the Women's Health Initiative hormone therapy trials. Arch Intern Med. 2010 Oct 11;170(18):1678-85. doi: 10.1001/archinternmed.2010.342. PMID 20937929
- [Derived] Rajpathak SN, Xue X, Wassertheil-Smoller S, Van Horn L, Snetselaar L, Martin LW, Rohan TE. Effect of long term low-fat dietary intervention on change in hemostatic factors: results from the Women's Health Initiative. Nutr Metab Cardiovasc Dis. 2012 Apr;22(4):337-9. doi: 10.1016/j.numecd.2010.07.002. Epub 2010 Sep 29. PMID 20884191
- [Derived] Chlebowski RT, Menon R, Chaisanguanthum RM, Jackson DM. Prospective evaluation of two recruitment strategies for a randomized controlled cancer prevention trial. Clin Trials. 2010 Dec;7(6):744-8. doi: 10.1177/1740774510383886. Epub 2010 Sep 10. PMID 20833684
- [Derived] Prentice RL, Paczesny S, Aragaki A, Amon LM, Chen L, Pitteri SJ, McIntosh M, Wang P, Buson Busald T, Hsia J, Jackson RD, Rossouw JE, Manson JE, Johnson K, Eaton C, Hanash SM. Novel proteins associated with risk for coronary heart disease or stroke among postmenopausal women identified by in-depth plasma proteome profiling. Genome Med. 2010 Jul 28;2(7):48. doi: 10.1186/gm169. PMID 20667078
- [Derived] Kuller LH, Margolis KL, Gaussoin SA, Bryan NR, Kerwin D, Limacher M, Wassertheil-Smoller S, Williamson J, Robinson JG; Women's Health Initiative Memory Study Research Group. Relationship of hypertension, blood pressure, and blood pressure control with white matter abnormalities in the Women's Health Initiative Memory Study (WHIMS)-MRI trial. J Clin Hypertens (Greenwich). 2010 Mar;12(3):203-12. doi: 10.1111/j.1751-7176.2009.00234.x. PMID 20433539
- [Derived] Robinson JG, Wallace R, Safford MM, Pettinger M, Cochrane B, Ko MG, O'Sullivan MJ, Masaki K, Petrovich H. Another treatment gap: restarting secondary prevention medications: the Women's Health Initiative. J Clin Lipidol. 2010 Jan-Feb;4(1):36-45. doi: 10.1016/j.jacl.2009.12.006. PMID 20354566
- [Derived] Rajpathak SN, Xue X, Wassertheil-Smoller S, Van Horn L, Robinson JG, Liu S, Allison M, Martin LW, Ho GY, Rohan TE. Effect of 5 y of calcium plus vitamin D supplementation on change in circulating lipids: results from the Women's Health Initiative. Am J Clin Nutr. 2010 Apr;91(4):894-9. doi: 10.3945/ajcn.2009.28579. Epub 2010 Feb 24. PMID 20181812
- [Derived] Hsia J, Rodabough RJ, Manson JE, Liu S, Freiberg MS, Graettinger W, Rosal MC, Cochrane B, Lloyd-Jones D, Robinson JG, Howard BV; Women's Health Initiative Research Group. Evaluation of the American Heart Association cardiovascular disease prevention guideline for women. Circ Cardiovasc Qual Outcomes. 2010 Mar;3(2):128-34. doi: 10.1161/CIRCOUTCOMES.108.842385. Epub 2010 Feb 16. PMID 20160160
- [Derived] Toh S, Hernandez-Diaz S, Logan R, Rossouw JE, Hernan MA. Coronary heart disease in postmenopausal recipients of estrogen plus progestin therapy: does the increased risk ever disappear? A randomized trial. Ann Intern Med. 2010 Feb 16;152(4):211-7. doi: 10.7326/0003-4819-152-4-201002160-00005. PMID 20157135
- [Derived] Prentice RL, Huang Y, Hinds DA, Peters U, Cox DR, Beilharz E, Chlebowski RT, Rossouw JE, Caan B, Ballinger DG. Variation in the FGFR2 gene and the effect of a low-fat dietary pattern on invasive breast cancer. Cancer Epidemiol Biomarkers Prev. 2010 Jan;19(1):74-9. doi: 10.1158/1055-9965.EPI-09-0663. PMID 20056625
- [Derived] Prentice RL, Huang Y, Hinds DA, Peters U, Pettinger M, Cox DR, Beilharz E, Chlebowski RT, Rossouw JE, Caan B, Ballinger DG. Variation in the FGFR2 gene and the effects of postmenopausal hormone therapy on invasive breast cancer. Cancer Epidemiol Biomarkers Prev. 2009 Nov;18(11):3079-85. doi: 10.1158/1055-9965.EPI-09-0611. Epub 2009 Oct 27. PMID 19861516
- [Derived] Crandall CJ, Aragaki AK, Chlebowski RT, McTiernan A, Anderson G, Hendrix SL, Cochrane BB, Kuller LH, Cauley JA. New-onset breast tenderness after initiation of estrogen plus progestin therapy and breast cancer risk. Arch Intern Med. 2009 Oct 12;169(18):1684-91. doi: 10.1001/archinternmed.2009.303. PMID 19822825
- [Derived] Chlebowski RT, Schwartz AG, Wakelee H, Anderson GL, Stefanick ML, Manson JE, Rodabough RJ, Chien JW, Wactawski-Wende J, Gass M, Kotchen JM, Johnson KC, O'Sullivan MJ, Ockene JK, Chen C, Hubbell FA; Women's Health Initiative Investigators. Oestrogen plus progestin and lung cancer in postmenopausal women (Women's Health Initiative trial): a post-hoc analysis of a randomised controlled trial. Lancet. 2009 Oct 10;374(9697):1243-51. doi: 10.1016/S0140-6736(09)61526-9. Epub 2009 Sep 18. PMID 19767090
- [Derived] Kabat GC, Kim M, Adams-Campbell LL, Caan BJ, Chlebowski RT, Neuhouser ML, Shikany JM, Rohan TE; WHI Investigators. Longitudinal study of serum carotenoid, retinol, and tocopherol concentrations in relation to breast cancer risk among postmenopausal women. Am J Clin Nutr. 2009 Jul;90(1):162-9. doi: 10.3945/ajcn.2009.27568. Epub 2009 May 27. PMID 19474140
- [Derived] Prentice RL, Pettinger M, Beresford SA, Wactawski-Wende J, Hubbell FA, Stefanick ML, Chlebowski RT. Colorectal cancer in relation to postmenopausal estrogen and estrogen plus progestin in the Women's Health Initiative clinical trial and observational study. Cancer Epidemiol Biomarkers Prev. 2009 May;18(5):1531-7. doi: 10.1158/1055-9965.EPI-08-1209. PMID 19423530
- [Derived] McTiernan A, Wactawski-Wende J, Wu L, Rodabough RJ, Watts NB, Tylavsky F, Freeman R, Hendrix S, Jackson R; Women's Health Initiative Investigators. Low-fat, increased fruit, vegetable, and grain dietary pattern, fractures, and bone mineral density: the Women's Health Initiative Dietary Modification Trial. Am J Clin Nutr. 2009 Jun;89(6):1864-76. doi: 10.3945/ajcn.2008.26956. Epub 2009 Apr 29. PMID 19403636
- [Derived] Katayama H, Paczesny S, Prentice R, Aragaki A, Faca VM, Pitteri SJ, Zhang Q, Wang H, Silva M, Kennedy J, Rossouw J, Jackson R, Hsia J, Chlebowski R, Manson J, Hanash S. Application of serum proteomics to the Women's Health Initiative conjugated equine estrogens trial reveals a multitude of effects relevant to clinical findings. Genome Med. 2009 Apr 29;1(4):47. doi: 10.1186/gm47. PMID 19402886
- [Derived] LaCroix AZ, Kotchen J, Anderson G, Brzyski R, Cauley JA, Cummings SR, Gass M, Johnson KC, Ko M, Larson J, Manson JE, Stefanick ML, Wactawski-Wende J. Calcium plus vitamin D supplementation and mortality in postmenopausal women: the Women's Health Initiative calcium-vitamin D randomized controlled trial. J Gerontol A Biol Sci Med Sci. 2009 May;64(5):559-67. doi: 10.1093/gerona/glp006. Epub 2009 Feb 16. PMID 19221190
- [Derived] Neuhouser ML, Wassertheil-Smoller S, Thomson C, Aragaki A, Anderson GL, Manson JE, Patterson RE, Rohan TE, van Horn L, Shikany JM, Thomas A, LaCroix A, Prentice RL. Multivitamin use and risk of cancer and cardiovascular disease in the Women's Health Initiative cohorts. Arch Intern Med. 2009 Feb 9;169(3):294-304. doi: 10.1001/archinternmed.2008.540. PMID 19204221
- [Derived] Hsia J, Larson JC, Ockene JK, Sarto GE, Allison MA, Hendrix SL, Robinson JG, LaCroix AZ, Manson JE; Women's Health Initiative Research Group. Resting heart rate as a low tech predictor of coronary events in women: prospective cohort study. BMJ. 2009 Feb 3;338:b219. doi: 10.1136/bmj.b219. PMID 19193613
- [Derived] Thomson CA, Neuhouser ML, Shikany JM, Caan BJ, Monk BJ, Mossavar-Rahmani Y, Sarto G, Parker LM, Modugno F, Anderson GL. The role of antioxidants and vitamin A in ovarian cancer: results from the Women's Health Initiative. Nutr Cancer. 2008;60(6):710-9. doi: 10.1080/01635580802233983. PMID 19005970
- [Derived] Rossouw JE, Cushman M, Greenland P, Lloyd-Jones DM, Bray P, Kooperberg C, Pettinger M, Robinson J, Hendrix S, Hsia J. Inflammatory, lipid, thrombotic, and genetic markers of coronary heart disease risk in the women's health initiative trials of hormone therapy. Arch Intern Med. 2008 Nov 10;168(20):2245-53. doi: 10.1001/archinte.168.20.2245. PMID 19001202
- [Derived] Tinker LF, Bonds DE, Margolis KL, Manson JE, Howard BV, Larson J, Perri MG, Beresford SA, Robinson JG, Rodriguez B, Safford MM, Wenger NK, Stevens VJ, Parker LM; Women's Health Initiative. Low-fat dietary pattern and risk of treated diabetes mellitus in postmenopausal women: the Women's Health Initiative randomized controlled dietary modification trial. Arch Intern Med. 2008 Jul 28;168(14):1500-11. doi: 10.1001/archinte.168.14.1500. PMID 18663162
- [Derived] Zheng Z, Margolis KL, Liu S, Tinker LF, Ye W; Women's Health Initiative Investigators. Effects of estrogen with and without progestin and obesity on symptomatic gastroesophageal reflux. Gastroenterology. 2008 Jul;135(1):72-81. doi: 10.1053/j.gastro.2008.03.039. Epub 2008 Mar 25. PMID 18502208
- [Derived] Bray PF, Larson JC, Lacroix AZ, Manson J, Limacher MC, Rossouw JE, Lasser NL, Lawson WE, Stefanick ML, Langer RD, Margolis KL; Women's Health Initiative Investigators. Usefulness of baseline lipids and C-reactive protein in women receiving menopausal hormone therapy as predictors of treatment-related coronary events. Am J Cardiol. 2008 Jun 1;101(11):1599-1605. doi: 10.1016/j.amjcard.2008.01.043. Epub 2008 Apr 2. PMID 18489937
- [Derived] Heiss G, Wallace R, Anderson GL, Aragaki A, Beresford SA, Brzyski R, Chlebowski RT, Gass M, LaCroix A, Manson JE, Prentice RL, Rossouw J, Stefanick ML; WHI Investigators. Health risks and benefits 3 years after stopping randomized treatment with estrogen and progestin. JAMA. 2008 Mar 5;299(9):1036-45. doi: 10.1001/jama.299.9.1036. PMID 18319414
- [Derived] Chlebowski RT, Anderson G, Pettinger M, Lane D, Langer RD, Gilligan MA, Walsh BW, Chen C, McTiernan A; Women's Health Initiative Investigators. Estrogen plus progestin and breast cancer detection by means of mammography and breast biopsy. Arch Intern Med. 2008 Feb 25;168(4):370-7; quiz 345. doi: 10.1001/archinternmed.2007.123. PMID 18299491
- [Derived] de Boer IH, Tinker LF, Connelly S, Curb JD, Howard BV, Kestenbaum B, Larson JC, Manson JE, Margolis KL, Siscovick DS, Weiss NS; Women's Health Initiative Investigators. Calcium plus vitamin D supplementation and the risk of incident diabetes in the Women's Health Initiative. Diabetes Care. 2008 Apr;31(4):701-7. doi: 10.2337/dc07-1829. Epub 2008 Jan 30. PMID 18235052
- [Derived] Prentice RL, Thomson CA, Caan B, Hubbell FA, Anderson GL, Beresford SA, Pettinger M, Lane DS, Lessin L, Yasmeen S, Singh B, Khandekar J, Shikany JM, Satterfield S, Chlebowski RT. Low-fat dietary pattern and cancer incidence in the Women's Health Initiative Dietary Modification Randomized Controlled Trial. J Natl Cancer Inst. 2007 Oct 17;99(20):1534-43. doi: 10.1093/jnci/djm159. Epub 2007 Oct 9. PMID 17925539
- [Derived] Manson JE, Allison MA, Rossouw JE, Carr JJ, Langer RD, Hsia J, Kuller LH, Cochrane BB, Hunt JR, Ludlam SE, Pettinger MB, Gass M, Margolis KL, Nathan L, Ockene JK, Prentice RL, Robbins J, Stefanick ML; WHI and WHI-CACS Investigators. Estrogen therapy and coronary-artery calcification. N Engl J Med. 2007 Jun 21;356(25):2591-602. doi: 10.1056/NEJMoa071513. PMID 17582069
- [Derived] Caan B, Neuhouser M, Aragaki A, Lewis CB, Jackson R, LeBoff MS, Margolis KL, Powell L, Uwaifo G, Whitlock E, Wylie-Rosett J, LaCroix A. Calcium plus vitamin D supplementation and the risk of postmenopausal weight gain. Arch Intern Med. 2007 May 14;167(9):893-902. doi: 10.1001/archinte.167.9.893. PMID 17502530
- [Derived] Rossouw JE, Prentice RL, Manson JE, Wu L, Barad D, Barnabei VM, Ko M, LaCroix AZ, Margolis KL, Stefanick ML. Postmenopausal hormone therapy and risk of cardiovascular disease by age and years since menopause. JAMA. 2007 Apr 4;297(13):1465-77. doi: 10.1001/jama.297.13.1465. PMID 17405972
- [Derived] Denes P, Larson JC, Lloyd-Jones DM, Prineas RJ, Greenland P. Major and minor ECG abnormalities in asymptomatic women and risk of cardiovascular events and mortality. JAMA. 2007 Mar 7;297(9):978-85. doi: 10.1001/jama.297.9.978. PMID 17341712
- [Derived] Wactawski-Wende J, Kotchen JM, Anderson GL, Assaf AR, Brunner RL, O'Sullivan MJ, Margolis KL, Ockene JK, Phillips L, Pottern L, Prentice RL, Robbins J, Rohan TE, Sarto GE, Sharma S, Stefanick ML, Van Horn L, Wallace RB, Whitlock E, Bassford T, Beresford SA, Black HR, Bonds DE, Brzyski RG, Caan B, Chlebowski RT, Cochrane B, Garland C, Gass M, Hays J, Heiss G, Hendrix SL, Howard BV, Hsia J, Hubbell FA, Jackson RD, Johnson KC, Judd H, Kooperberg CL, Kuller LH, LaCroix AZ, Lane DS, Langer RD, Lasser NL, Lewis CE, Limacher MC, Manson JE; Women's Health Initiative Investigators. Calcium plus vitamin D supplementation and the risk of colorectal cancer. N Engl J Med. 2006 Feb 16;354(7):684-96. doi: 10.1056/NEJMoa055222. PMID 16481636
- See also: Related Info — http://www.nhlbi.nih.gov/whi/